CLINICAL TRIAL: NCT03387813
Title: Hemodynamic-GUIDEd Management of Heart Failure
Acronym: GUIDE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIP-10170
Record Dates: First submitted 2017-12-12; First posted 2018-01-02 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Heart Failure, Systolic; Heart Failure, Diastolic; Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure NYHA Class IV; Heart Failure，Congestive; Heart Failure With Reduced Ejection Fraction; Heart Failure With Normal Ejection Fraction; Heart Failure; With Decompensation
Keywords: Heart Failure; Hemodynamic Monitoring; CardioMEMS; Pulmonary Artery Pressure
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Heart Failure, Diastolic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Randomized Arm - Treatment Group (Experimental): Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  Interventions: Device: CardioMEMS™ HF System
- Randomized Arm - Control Group (Experimental): Management of subjects per standard of care (signs, symptoms, weight etc.) without knowledge of PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  Interventions: Device: CardioMEMS™ HF System
- Single Arm (Experimental): Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  Interventions: Device: CardioMEMS™ HF System

INTERVENTIONS:
Device: CardioMEMS™ HF System — The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Other Names: CardioMEMS; CardioMEMS PA Sensor; CardioMEMS HF System

SUMMARY:
The GUIDE-HF IDE clinical trial is intended to demonstrate the effectiveness of the CardioMEMS™ HF System in an expanded patient population including heart failure (HF) patients outside of the present indication, but at risk for future HF events or mortality.

DETAILED DESCRIPTION:
The GUIDE-HF IDE clinical trial is intended to demonstrate the effectiveness of the CardioMEMS™ HF System in an expanded patient population including HF patients outside of the present indication, but at risk for future HF events or mortality.

The trial includes patients with New York Heart Association (NYHA) Class II, III, or IV HF who have an elevated N-terminal pro-Brain Natriuretic Peptide (NT-proBNP) (or an elevated Brain Natriuretic Peptide (BNP)) and/or a prior HF hospitalization (HFH).

The GUIDE-HF IDE trial will include approximately 3600 subjects at approximately 140 North American sites and consists of two arms: a Randomized Arm and a Single Arm.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis and treatment for heart failure (HF) (regardless of left ventricular ejection fraction (LVEF)) for > 90 days prior to the date of consent:

   a. Subjects should be on stable, optimally titrated medical therapy for at least 30 days, as recommended according to current American Heart Association (AHA)/American College of Cardiology (ACC) guidelines as standard-of-care for HF therapy in the United States, with any intolerance documented.
2. GUIDE-HF Randomized Arm Only: NYHA Class II, III or IV HF symptoms documented within 30 days prior to consent.
3. GUIDE-HF Single Arm Only: NYHA Class III HF symptoms documented within 30 days prior to consent.
4. HF hospitalization (HFH) within 12 months prior to consent and/or elevated N-terminal pro-Brain Natriuretic Peptide (NT-proBNP) (or Brain Natriuretic Peptide (BNP)) within 30 days prior to consent defined as:

   1. Subjects with LVEF ≤ 40%: NT-proBNP ≥ 1000 pg/mL (or BNP ≥ 250 pg/mL).
   2. Subjects with LVEF > 40%: NT-proBNP ≥ 700 pg/mL (or BNP ≥ 175 pg/mL).
   3. Thresholds for NT-proBNP and BNP (for both LVEF ≤ 40% and LVEF > 40%) will be corrected for body mass index (BMI) using a 4% reduction per BMI unit over 25 kg/m2
5. ≥ 18 years of age
6. Chest circumference of < 65 inches, if BMI is > 35 kg/m2
7. Written informed consent obtained from subject
8. Willing and able to upload pulmonary artery (PA) pressure information and comply with the follow-up requirements

Exclusion Criteria:

1. Intolerance to all neuro-hormonal antagonists (i.e., intolerance to angiotensin converting enzyme-inhibitors (ACE-I), angiotensin receptor blockers (ARB), angiotensin-neprilysin inhibitors (ARNi), hydralazine/isosorbide dinitrate and beta-blockers)
2. ACC/AHA Stage D refractory HF (including having received or currently receiving pharmacologic circulatory support with inotropes)
3. Received or are likely to receive an advanced therapy (e.g., mechanical circulatory support or cardiac transplant) in the next 12 months
4. NYHA Class IV HF patients with:

   1. Continuous or chronic use of scheduled intermittent inotropic therapy for HF and an INTERMACS level of ≤ 4, OR
   2. Persistence of fluid overload with maximum (or dose equivalent) diuretic intervention
5. Glomerular Filtration Rate (eGFR) < 25 mL/min and non-responsive to diuretic therapy, or receiving chronic dialysis
6. Inability to tolerate or receive dual antiplatelet therapy or anticoagulation therapy for one month post-implantation
7. Significant congenital heart disease that has not been repaired and would prevent implantation of the CardioMEMS™ PA Sensor
8. Implanted with mechanical right heart valve(s)
9. Unrepaired severe valvular disease
10. Pregnant or planning to become pregnant in the next 12 months
11. An active, ongoing infection, defined as being febrile, an elevated white blood cell count, on intravenous antibiotics, and/or positive cultures (blood, sputum or urine).
12. History of current or recurrent (≥ 2 episodes within 5 years prior to consent) pulmonary emboli and/or deep vein thrombosis
13. Major cardiovascular event (e.g., unstable angina, myocardial infarction, percutaneous coronary intervention, open heart surgery, or stroke, etc.) within 90 days prior to consent
14. Implanted with Cardiac Resynchronization Therapy (CRT)-Pacemaker (CRT-P) or CRT-Defibrillator (CRT-D) for less than 90 days prior to consent
15. Enrollment into another trial with an active treatment arm
16. Anticipated life expectancy of < 12 months
17. Any condition that, in the opinion of the Investigator, would not allow for utilization of the CardioMEMS™ HF System to manage the subject using information gained from hemodynamic measurements to adjust medications, including the presence of unexpectedly severe pulmonary hypertension (e.g., trans-pulmonary gradient >15) at implant right heart catheterization (RHC), a history of non-compliance, or any condition that would preclude CardioMEMS™ PA Sensor implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2358 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nessa Johnson, PhD, Study Director — Abbott
Locations (129):
- United States (125):
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - John Muir Medical Center, Concord, California
  - Adventist Health St. Helena, Deer Park, California
  - Scripps Health, La Jolla, California
  - University of California at San Diego (UCSD) Medical Center, La Jolla, California
  - USC University Hospital, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Sutter Medical Center, Sacramento, Sacramento, California
  - Mercy Medical Group - Cardiology, Sacramento, California
  - San Diego Cardiac Center, San Diego, California
  - California Pacific Medical Center - Van Ness Campus, San Francisco, California
  - Ventura Cardiology Consultants, Ventura, California
  - University of Colorado Hospital, Aurora, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Bethesda Memorial Hospital, Boynton Beach, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Advent Health Orlando, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Athens Regional Medical Center, Athens, Georgia
  - University Hospital, Augusta, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Northshore University HealthSystem, Evanston, Illinois
  - Advocate Health and Hospitals Corporation, Oakbrook Terrace, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Heart Center of Lake County, Merrillville, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Our Lady of the Lake Hospital, Baton Rouge, Louisiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Advanced Cardiovascular Specialists, Shreveport, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - McLaren Health Care Corporation, Auburn Hills, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - MidMichigan Medical Center-Midland, Midland, Michigan
  - Providence Hospital, Southfield, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - BryanLGH Heart Institute, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Catholic Medical Center, Manchester, New Hampshire
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - New York University Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - New York-Presbyterian/Columbia University, New York, New York
  - Hudson Valley Cardiovascular Practice, P.C., Poughkeepsie, New York
  - Rochester General Hospital, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - WakeMed Hospital, Raleigh, North Carolina
  - Akron City Hospital, Akron, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - St. Elizabeth Health Center, Youngstown, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital South, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute at Utica, Tulsa, Oklahoma
  - Providence Heart and Vascular, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Pinnacle Health System, Harrisburg, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital - ASRI, Pittsburgh, Pennsylvania
  - The Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Main Line Health Center/Lankenau Hospital, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health-Midlands, Columbia, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - St Thomas Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Acension Texas Cardiovascular, Austin, Texas
  - Austin Heart, Austin, Texas
  - Baylor University Hospital, Dallas, Texas
  - John Peter Smith Hospital, Fort Worth, Texas
  - Park Plaza Hospital, Houston, Texas
  - CHI St. Luke's Health Baylor College of Medicine Med. Ctr., Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - Virginia Heart - The Cardiovascular Group, P.C., Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Bon Secours Heart & Vascular Institute, Richmond, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Providence Everett Medical Center, Everett, Washington
  - Swedish Medical Center - Heart & Vascular, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Aurora Medical Group, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Wausau Hospital, Wausau, Wisconsin
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - Vancouver General Hospital (U of BC), Vancouver, British Columbia
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zile MR, Abraham WT, Stevenson LW, Costanzo MR, Angermann CE, Mehra MR, Desai AS, Ducharme A, Johnson N, Henderson J, Lindenfeld J. Relationship Between Remote, Ambulatory Pulmonary Artery Pressures, and All-Cause Mortality in Patients With Chronic Heart Failure. Circ Heart Fail. 2025 Jun;18(6):e012754. doi: 10.1161/CIRCHEARTFAILURE.124.012754. Epub 2025 Apr 14. PMID 40223608
- [Derived] Desai AS, Maisel A, Mehra MR, Zile MR, Ducharme A, Paul S, Sears SF, Smart F, Bhatt K, Krim S, Henderson J, Johnson N, Adamson PB, Costanzo MR, Lindenfeld J; GUIDE-HF Investigators. Hemodynamic-Guided Heart Failure Management in Patients With Either Prior HF Hospitalization or Elevated Natriuretic Peptides. JACC Heart Fail. 2023 Jun;11(6):691-698. doi: 10.1016/j.jchf.2023.01.007. Epub 2023 Apr 12. PMID 37286262
- [Derived] Zile MR, Mehra MR, Ducharme A, Sears SF, Desai AS, Maisel A, Paul S, Smart F, Grafton G, Kumar S, Nossuli TO, Johnson N, Henderson J, Adamson PB, Costanzo MR, Lindenfeld J. Hemodynamically-Guided Management of Heart Failure Across the Ejection Fraction Spectrum: The GUIDE-HF Trial. JACC Heart Fail. 2022 Dec;10(12):931-944. doi: 10.1016/j.jchf.2022.08.012. Epub 2022 Oct 12. PMID 36456066
- [Derived] Zile MR, Desai AS, Costanzo MR, Ducharme A, Maisel A, Mehra MR, Paul S, Sears SF, Smart F, Chien C, Guha A, Guichard JL, Hall S, Jonsson O, Johnson N, Sood P, Henderson J, Adamson PB, Lindenfeld J. The GUIDE-HF trial of pulmonary artery pressure monitoring in heart failure: impact of the COVID-19 pandemic. Eur Heart J. 2022 Jul 14;43(27):2603-2618. doi: 10.1093/eurheartj/ehac114. PMID 35266003
- [Derived] Lindenfeld J, Zile MR, Desai AS, Bhatt K, Ducharme A, Horstmanshof D, Krim SR, Maisel A, Mehra MR, Paul S, Sears SF, Sauer AJ, Smart F, Zughaib M, Castaneda P, Kelly J, Johnson N, Sood P, Ginn G, Henderson J, Adamson PB, Costanzo MR. Haemodynamic-guided management of heart failure (GUIDE-HF): a randomised controlled trial. Lancet. 2021 Sep 11;398(10304):991-1001. doi: 10.1016/S0140-6736(21)01754-2. Epub 2021 Aug 27. PMID 34461042

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized Arm enrolled 1022 subjects across 118 sites, of which 1000 are endpoint-contributing (successfully implanted and randomized). Subject enrollment took place between March 2018 and December 2019, with the last follow-up completed in January 2021.
  Single Arm enrolled 1401 subjects across 119 sites, of which 1358 are endpoint-contributing (successfully implanted). Subject enrollment took place between March 2018 and April 2022, with the last follow-up completed in May 2023.
Pre-assignment Details: 22 subjects were not randomized in the Randomized Arm and 43 subjects were not assigned to the Single Arm due to unsuccessful implantation attempts.
Groups:
- Randomized Arm - Treatment Group: Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Randomized Arm - Control Group: Management of subjects per standard of care (signs, symptoms, weight etc.) without knowledge of PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm: Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Period: Overall Study
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group | Single Arm
Started | 497 (Successful Implant and Randomized) | 503 (Successful Implant and Randomized) | 1358 (Successful Implant)
Complete 6 Month Follow-Up | 467 | 469 | 1238
Completed (Completed 12 Month Follow-Up) | 432 | 422 | 1076
Not Completed | 65 | 81 | 282
Not completed — Death | 40 | 37 | 190
Not completed — Withdrawal by Subject | 9 | 19 | 32
Not completed — Lost to Follow-up | 3 | 9 | 15
Not completed — Non-Compliance | 6 | 6 | 31
Not completed — Subject In Hospice/Relocated/Severe COVID-19/On Transplant List/PI Discretion | 7 | 10 | 14

BASELINE CHARACTERISTICS:
Population: The endpoint-contributing population consists of patients who were successfully implanted.
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group | Single Arm | Total
Number analyzed (Participants) | 497 | 503 | 1358 | 2358
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (11.1) | 69.2 (11.0) | 70.5 (10.9) | 69.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 188 | 584 | 959
  Male | 310 | 315 | 774 | 1399
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 17 | 61 | 94
  Not Hispanic or Latino | 477 | 483 | 1283 | 2243
  Unknown or Not Reported | 4 | 3 | 14 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 4 | 6
  Asian | 0 | 1 | 12 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 3 | 3
  Black or African American | 86 | 93 | 188 | 367
  White | 403 | 404 | 1125 | 1932
  More than one race | 1 | 1 | 3 | 5
  Unknown or Not Reported | 6 | 3 | 23 | 32
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 32.9 (8.3) | 33.8 (8.4) | 34.0 (8.8) | 33.8 (8.7)
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) functional classification of HF symptoms is designed to subjectively quantify an individual's burden of congestive symptoms in order to provide specific medical and device interventions appropriate for the patient's condition.
  NYHA classifications are categorized as class I (no limitation of physical activity), class II (slight limitation of physical activity), class III (marked limitation of physical activity) to class IV (symptoms of heart failure at rest). The higher the class, the more severe the heart failure symptoms. Population: Data not available in 1 subject in Single Arm. Subject did not record NYHA class following reconsent.
  Participants
    number analyzed (Participants) | 497 | 503 | 1357 | 2357
    Class II | 146 | 150 | 0 | 296
    Class III | 322 | 328 | 1356 | 2006
    Class IV | 29 | 25 | 1 | 55
Medical History - Ischemic etiology [Count of Participants; unit: Participants] | 207 | 190 | 489 | 886
Medical History - Previous myocardial infarction [Count of Participants; unit: Participants] | 144 | 158 | 359 | 661
Medical History - Previous percutaneous coronary intervention [Count of Participants; unit: Participants] | 165 | 158 | 379 | 702
Medical History - Previous coronary artery bypass grafting [Count of Participants; unit: Participants] | 135 | 136 | 331 | 602
Medical History - Diabetes [Count of Participants; unit: Participants] | 243 | 261 | 685 | 1189
Medical History - Cerebrovascular accident [Count of Participants; unit: Participants] | 66 | 65 | 186 | 317
Medical History - Atrial flutter or fibrillation [Count of Participants; unit: Participants] | 300 | 291 | 844 | 1435
Treatment History - Previous cardiac resynchronization therapy [Count of Participants; unit: Participants] | 142 | 163 | 367 | 672
Treatment History - Previous implantation of defibrillator [Count of Participants; unit: Participants] | 213 | 205 | 457 | 875
Heart rate [Mean (Standard Deviation); unit: beats per minute (bpm)] | 73.8 (12.5) | 74.2 (12.3) | 74.2 (12.5) | 74.1 (12.5)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Data not available for 1 subject from Single Arm.
  mmHg
    number analyzed (Participants) | 497 | 503 | 1357 | 2357
    (all) | 121.6 (19.1) | 120.8 (18.1) | 120.7 (19) | 120.9 (18.8)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Data not available for 1 subject from Single Arm.
  mmHg
    number analyzed (Participants) | 497 | 503 | 1357 | 2357
    (all) | 69.2 (10.8) | 69.0 (10.8) | 67.7 (10.8) | 68.3 (10.8)
Left ventricular ejection fraction [Mean (Standard Deviation); unit: %] | 39.4 (17.3) | 40.7 (16.9) | 43.5 (17.0) | 42.0 (17.1)
Left ventricular ejection fraction > 40% [Count of Participants; unit: Participants] | 224 | 245 | 752 | 1221
Pulmonary artery (PA) systolic pressure [Mean (Standard Deviation); unit: mmHg] | 44.9 (13.9) | 45.2 (14.6) | 46.7 (15.1) | 46.0 (14.8)
PA Diastolic Pressure [Mean (Standard Deviation); unit: mmHg] | 18.9 (8.0) | 18.8 (7.7) | 19.7 (7.6) | 19.4 (7.7)
PA Mean Pressure [Mean (Standard Deviation); unit: mmHg] | 29.2 (9.5) | 29.4 (10.0) | 30.2 (9.7) | 29.8 (9.7)
Pulmonary capillary wedge pressure [Mean (Standard Deviation); unit: mmHg] — Population: Data not available in 2 subjects from Randomized Arm (Treatment Group) and 8 subjects from Single Arm.
  mmHg
    number analyzed (Participants) | 495 | 503 | 1350 | 2348
    (all) | 17.3 (8.0) | 17.6 (7.9) | 18.0 (7.5) | 17.8 (7.7)
Cardiac output [Mean (Standard Deviation); unit: L/min] | 4.83 (2.62) | 4.70 (1.46) | 4.80 (1.55) | 4.78 (1.81)
Cardiac index [Mean (Standard Deviation); unit: L/min/m2] | 2.27 (1.11) | 2.19 (0.63) | 2.24 (0.66) | 2.24 (0.77)
Ambulatory Hemodynamics during First Week [Mean (Standard Deviation); unit: mmHg] — Ambulatory hemodynamics during the first week are pulmonary artery pressure readings collected from the CardioMEMS sensor during the initial week following its implantation. These readings serve as baseline measurements rather than study outcomes, as hemodynamic data can only be gathered using the CardioMEMS sensor post-implantation. Population: Data not available for 4 subjects in Randomized Arm (Control Group) and 8 subjects in Single Arm.
  mmHg
    PA Systolic Pressure: number analyzed (Participants) | 497 | 499 | 1350 | 2346
    PA Systolic Pressure | 46.3 (14.4) | 46.2 (13.3) | 47.4 (13.9) | 46.9 (13.9)
    PA Diastolic Pressure: number analyzed (Participants) | 497 | 499 | 1350 | 2346
    PA Diastolic Pressure | 22.4 (7.8) | 22.7 (7.4) | 23.0 (7.4) | 22.8 (7.5)
    PA Mean Pressure: number analyzed (Participants) | 497 | 499 | 1350 | 2346
    PA Mean Pressure | 31.8 (10.2) | 31.9 (9.6) | 32.6 (9.7) | 32.3 (9.8)
Ambulatory Heart Rate during First Week [Mean (Standard Deviation); unit: beats per minute (bpm)] — Ambulatory heart rate during the first week are heart rate readings collected from the CardioMEMS sensor during the initial week following its implantation. These readings serve as baseline measurements rather than study outcomes, as these measurements can only be gathered using the CardioMEMS sensor post-implantation. Population: Data not available in 4 subjects from Randomized Arm (Control Group) and 8 subjects in Single Arm.
  beats per minute (bpm)
    number analyzed (Participants) | 497 | 499 | 1350 | 2346
    (all) | 78.8 (11.7) | 79.4 (11.9) | 79.3 (11.9) | 79.2 (11.8)
Laboratory Analyses - Serum creatinine level [Mean (Standard Deviation); unit: μmol/L] — Population: Data not available in 2 subjects from Randomized Arm (Treatment Group), 8 subjects from Randomized (Control Group) and 5 subjects from Single Arm.
  μmol/L
    number analyzed (Participants) | 495 | 495 | 1353 | 2343
    (all) | 128.5 (44.5) | 133.5 (48.5) | 134.1 (49.4) | 132.8 (48.2)
Laboratory Analyses - Estimated glomerular filtration rate [Mean (Standard Deviation); unit: ml/min/1.73m2] — Population: Data not available for 2 subjects from Randomized Arm (Treatment Group), 9 subjects from Randomized Arm (Control Group) and 5 subjects from Single Arm.
  ml/min/1.73m2
    number analyzed (Participants) | 495 | 494 | 1353 | 2342
    (all) | 54.3 (21.3) | 52.8 (20.8) | 51.2 (21.3) | 52.2 (21.2)
Laboratory Analyses - Brain Natriuretic Peptide (BNP) [Mean (Standard Deviation); unit: pg/mL] — Population: Data not available for 236 subjects from Randomized Arm (Treatment Group), 247 subjects from Randomized Arm (Control Group) and 688 subjects from Single Arm.
  pg/mL
    number analyzed (Participants) | 261 | 256 | 670 | 1187
    (all) | 520.7 (689.2) | 552.4 (954) | 517 (618.8) | 525.4 (718.3)
Laboratory Analyses - N-terminal pro-B-type natriuretic peptide (NT-proBNP) [Mean (Standard Deviation); unit: pg/mL] — Population: Data not available for 278 subjects from Randomized Arm (Treatment Group), 278 subjects from Randomized Arm (Control Group) and 715 subjects from Single Arm.
  pg/mL
    number analyzed (Participants) | 219 | 225 | 643 | 1087
    (all) | 2460 (3707) | 2183 (2803) | 2446 (3521) | 2395 (3423)
ACE-Inhibitor or ARB or ARNi [Count of Participants; unit: Participants] | 319 | 320 | 702 | 1341
ARNi [Count of Participants; unit: Participants] | 145 | 139 | 318 | 602
Beta Blocker [Count of Participants; unit: Participants] | 444 | 442 | 1126 | 2012
Mineralocorticoid Receptor Antagonist [Count of Participants; unit: Participants] | 237 | 216 | 613 | 1066
Diuretic [Count of Participants; unit: Participants] | 474 | 478 | 1322 | 2274
Hydralazine [Count of Participants; unit: Participants] | 81 | 80 | 200 | 361
Nitrate [Count of Participants; unit: Participants] | 99 | 103 | 246 | 448
SGLT2 Inhibitor [Count of Participants; unit: Participants] — Population: Data not available for 345 subjects from Randomized Arm (Treatment Group), 363 subjects from Randomized Arm (Control Group) and 363 subjects from Single Arm.
  Participants
    number analyzed (Participants) | 152 | 140 | 995 | 1287
    (all) | 2 | 2 | 115 | 119
Enrollment Type - Prior Heart Failure Hospitalization Only [Count of Participants; unit: Participants] — Population: One subject from Randomized Arm (Control Group) was enrolled and randomized but did not meet entry criteria for either a prior HFH or elevated NT-proBNP or BNP.
  Fourteen (14) subjects from the Single Arm were enrolled and implanted successfully but did not meet entry criteria for either a prior HFH or elevated NT-proBNP or BNP.
  Participants
    number analyzed (Participants) | 497 | 502 | 1344 | 2343
    (all) | 170 | 191 | 549 | 910
Enrollment Type - Prior Elevated NT-proBNP/BNP [Count of Participants; unit: Participants] — Population: One subject from Randomized Arm (Control Group) was enrolled and randomized but did not meet entry criteria for either a prior HFH or elevated NT-proBNP or BNP.
  Fourteen (14) subjects from the Single Arm were enrolled and implanted successfully but did not meet entry criteria for either a prior HFH or elevated NT-proBNP or BNP.
  Participants
    number analyzed (Participants) | 497 | 502 | 1344 | 2343
    (all) | 230 | 212 | 452 | 894
Enrollment Type - Prior Heart Failure Hospitalization and Elevated NT-proBNP/BNP [Count of Participants; unit: Participants] — Population: One subject from Randomized Arm (Control Group) was enrolled and randomized but did not meet entry criteria for either a prior HFH or elevated NT-proBNP or BNP.
  Fourteen (14) subjects from the Single Arm were enrolled and implanted successfully but did not meet entry criteria for either a prior HFH or elevated NT-proBNP or BNP.
  Participants
    number analyzed (Participants) | 497 | 502 | 1344 | 2343
    (all) | 97 | 99 | 343 | 539
KCCQ-12 Score [Mean (Standard Deviation); unit: scores on a scale] — The Kansas City Cardiomyopathy Questionnaire (KCCQ-12) is a validated health-related quality of life measure for heart failure and was qualified by the FDA as a medical device development tool in 2017. The KCCQ-12 quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life over a scale from 0 to 100. An overall summary score (OSS) is derived by averaging scores from each domain, with a higher score reflecting a better health status. Population: Data not available for 3 subjects from Randomized Arm (Treatment Group), 6 subjects from Randomized Arm (Control Group) and 7 subjects from Single Arm.
  scores on a scale
    number analyzed (Participants) | 494 | 497 | 1351 | 2342
    (all) | 54.9 (24.3) | 54.9 (23.8) | 48.8 (22.3) | 51.4 (23.2)
6-minute Walk Test (6MHW) [Mean (Standard Deviation); unit: meters] — Population: Data not available for 23 subjects from Randomized Arm (Treatment Group), 21 subjects from Randomized Arm (Control Group) and 101 subjects from Single Arm.
  meters
    number analyzed (Participants) | 474 | 482 | 1257 | 2213
    (all) | 235.2 (120.2) | 229.6 (123.0) | 196.9 (127.4) | 212.2 (126.2)

OUTCOME MEASURES:

1. Primary Outcome: (Randomized Arm) Composite Outcome of (1) HFHs, (2) Intravenous Diuretic Visits, and (3) All-cause Mortality
Description: The composite of:
  1. The number of recurrent heart failure hospitalizations (HFHs)
  2. The number of heart failure (HF) emergency department/hospital outpatient observation visits for intravenous diuretic therapy (ED/OP)
  3. The number of deaths of any cause
  added together with equal weighting into a total number of events
Time Frame: 12 months post-implantation (395 days after implant date)
Population: The primary endpoint was analyzed in the endpoint-contributing population, which included subjects that were successfully implanted and randomized.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 497 | 503
events per patient-year | 0.563 | 0.640
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group vs Randomized Arm - Control Group; Test type: Superiority; p = 0.1624, Anderson-Gill model (robust sandwich); Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.74 to 1.05]

2. Primary Outcome: (Randomized Arm) Composite Outcome of (1) HFHs, (2) Intravenous Diuretic Visits, and (3) All-cause Mortality [Follow-up Based COVID-19 Sensitivity Analysis]
Description: as for outcome 1
Time Frame: The COVID-19 pandemic occurred during follow-up after enrollment of all subjects. Events were analyzed through March 13, 2020 for pre-COVID-19 (median follow-up: 8.4 months) and after March 13, 2020 for during COVID-19 (median follow-up: 5.2 months).
Population: The primary endpoint limited to the follow-up period occurring "Pre-COVID-19" or "During COVID-19" was analyzed in the endpoint-contributing population including subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. All subjects were assessed based on their follow-up time occurring pre- or during-COVID periods using a time-varying covariate in the Andersen-Gill model. The Arm/Group Titles represent the follow-up time period.
Measure: Number; unit: events per patient-year
Groups:
- Randomized Arm - Treatment Group [Pre-COVID-19]; Randomized Arm - Treatment Group [During COVID-19]: Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Randomized Arm - Control Group [Pre-COVID-19]; Randomized Arm - Control Group [During COVID-19]: Management of subjects per standard of care (signs, symptoms, weight etc.) without knowledge of PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Randomized Arm - Treatment Group [Pre-COVID-19] | Randomized Arm - Control Group [Pre-COVID-19] | Randomized Arm - Treatment Group [During COVID-19] | Randomized Arm - Control Group [During COVID-19]
Number analyzed (Participants) | 497 | 503 | 497 | 503
events per patient-year | 0.553 | 0.682 | 0.597 | 0.536

3. Primary Outcome: (Randomized Arm) Composite Outcome of (1) HFHs, (2) Intravenous Diuretic Visits, and (3) All-cause Mortality [Subject Based COVID-19 Sensitivity Analysis]
Description: as for outcome 1
Time Frame: 12 Months Post Implantation
Population: The primary endpoint was analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Number; unit: events per patient-year
Groups:
- Randomized Arm - Treatment Group (Pre-COVID-19): Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending prior to COVID-19.
- Randomized Arm - Control Group (Pre-COVID-19): Management of subjects per standard of care (signs, symptoms, weight etc.) without knowledge of PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending prior to COVID-19.
- Randomized Arm - Treatment Group (During COVID-19): Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending during COVID-19.
- Randomized Arm - Control Arm (During COVID-19): Management of subjects per standard of care (signs, symptoms, weight etc.) without knowledge of PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending during COVID-19.
Arm/Group | Randomized Arm - Treatment Group (Pre-COVID-19) | Randomized Arm - Control Group (Pre-COVID-19) | Randomized Arm - Treatment Group (During COVID-19) | Randomized Arm - Control Arm (During COVID-19)
Number analyzed (Participants) | 187 | 196 | 310 | 307
events per patient-year | 0.710 | 0.864 | 0.508 | 0.539

4. Primary Outcome: (Randomized Arm) Composite Outcome of (1) HFHs, (2) Intravenous Diuretic Visits, and (3) All-cause Mortality [Event Based COVID-19 Sensitivity Analysis]
Description: as for outcome 1
Time Frame: 12 Months Post-Implantation
Population: The primary endpoint was analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. All subjects were enrolled before COVID-19 period (March 13, 2020). The event based COVID-19 sensitivity analysis compares treatment effect by excluding events adjudicated as either related or possible related to COVID-19.
Measure: Number; unit: events per patient-year
Groups:
- Randomized Arm - Treatment Group [Excluding COVID-19 Related Events]; Randomized Arm - Treatment Group [Excluding COVID-19 Related or Possibly Related Events]: Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Randomized Arm - Control Group [Excluding COVID-19 Related Events]; Randomized Arm - Control Group [Excluding COVID-19 Related or Possibly Related Events]: Management of subjects per standard of care (signs, symptoms, weight etc.) without knowledge of PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Randomized Arm - Treatment Group [Excluding COVID-19 Related Events] | Randomized Arm - Control Group [Excluding COVID-19 Related Events] | Randomized Arm - Treatment Group [Excluding COVID-19 Related or Possibly Related Events] | Randomized Arm - Control Group [Excluding COVID-19 Related or Possibly Related Events]
Number analyzed (Participants) | 497 | 503 | 497 | 503
events per patient-year | 0.563 | 0.633 | 0.558 | 0.619

5. Primary Outcome: (Single Arm) Composite Outcome of (1) HFHs, (2) Intravenous Diuretic Visits, and (3) All-cause Mortality
Description: The composite outcome of:
  1. The number of recurrent heart failure hospitalizations (HFHs)
  2. The number of emergency department/hospital outpatient observation visits for intravenous diuretic therapy
  3. The number of deaths of any cause
  added together with equal weighting into a total number of events
Time Frame: 12 months post-implantation (395 days after implant date)
Population: The primary endpoint was compared between subjects in the qualifying with elevated NT-proBNP/BNP levels only group and subjects in the qualifying with prior HF hospitalization only group.
Measure: Number; unit: events per patient-year
Groups:
- Single Arm - Elevated NT-proBNP/BNP Only: All subjects had prior elevated NT-proBNP/BNP only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm - Previous HF Hospitalization Only: All subjects had prior HF hospitalization only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only
Number analyzed (Participants) | 452 | 549
events per patient-year | 0.394 | 0.771
Statistical Analysis 1: Comparison: Single Arm - Elevated NT-proBNP/BNP Only vs Single Arm - Previous HF Hospitalization Only; Test type: Equivalence — Clinical equivalence was met if the lower limit of the confidence interval (CI) of ln(HR) for the primary endpoint in Elevated NT-proBNP/BNP only vs. prior HFH only subjects is > -0.2877 and the upper limit is < 0.2877; Hazard Ratio (HR) = 0.51, 90% CI 2-sided [0.44 to 0.60]

6. Primary Outcome: (Single Arm) Composite Outcome of (1) HFHs, (2) Intravenous Diuretic Visits, and (3) All-cause Mortality [Follow-up Based COVID-19 Sensitivity Analysis]
Description: as for outcome 5
Time Frame: Events were analyzed through March 13, 2020 for pre-COVID-19 analysis (median follow-up: 5.4 months) and from March 13, 2020 through the end of subject's follow-up for during COVID-19 analysis (median follow-up: 11.2 months).
Population: The primary endpoint limited to the follow-up period occurring "Prior to COVID-19" or "During COVID-19" was compared between subjects in the qualifying with elevated NT-proBNP/BNP levels only group and subjects in the qualifying with prior HF hospitalization only group. Subjects were assessed based on their follow-up time occurring pre- or during-COVID periods using a time-varying covariate. The Arm/Group Titles represent the follow-up time period.
Measure: Number; unit: events per patient-year
Groups:
- Single Arm - Elevated NT-proBNP/BNP Only [Prior to COVID-19]; Single Arm - Elevated NT-proBNP/BNP Only [During COVID-19]: All subjects had prior elevated NT-proBNP/BNP only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm - Previous HF Hospitalization Only [Prior to COVID-19]; Single Arm - Previous HF Hospitalization Only [During COVID-19]: All subjects had prior HF hospitalization only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Prior to COVID-19] | Single Arm - Previous HF Hospitalization Only [Prior to COVID-19] | Single Arm - Elevated NT-proBNP/BNP Only [During COVID-19] | Single Arm - Previous HF Hospitalization Only [During COVID-19]
Number analyzed (Participants) | 452 | 549 | 452 | 549
events per patient-year | 0.263 | 0.861 | 0.418 | 0.744

7. Primary Outcome: (Single Arm) Composite Outcome of (1) HFHs, (2) Intravenous Diuretic Visits, and (3) All-cause Mortality [Subject Based COVID-19 Sensitivity Analysis]
Description: as for outcome 5
Time Frame: 12 Months Post Implantation
Population: The primary endpoint was compared between subjects in the qualifying with elevated NT-proBNP/BNP levels only group and subjects in the qualifying with prior HF hospitalization only group. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Number; unit: events per patient-year
Groups:
- Single Arm - Elevated NT-proBNP/BNP Only (Pre-COVID-19); Single Arm - Elevated NT-proBNP/BNP Only (During COVID-19): All subjects had prior elevated NT-proBNP/BNP only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm - Previous HF Hospitalization Only (Pre-COVID-19); Single Arm - Previous HF Hospitalization Only (During COVID-19): All subjects had prior HF hospitalization only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only (Pre-COVID-19) | Single Arm - Previous HF Hospitalization Only (Pre-COVID-19) | Single Arm - Elevated NT-proBNP/BNP Only (During COVID-19) | Single Arm - Previous HF Hospitalization Only (During COVID-19)
Number analyzed (Participants) | 25 | 69 | 427 | 480
events per patient-year | 0.582 | 1.853 | 0.391 | 0.698

8. Primary Outcome: (Single Arm) Composite Outcome of (1) HFHs, (2) Intravenous Diuretic Visits, and (3) All-cause Mortality [Event Based COVID-19 Sensitivity Analysis]
Description: as for outcome 5
Time Frame: 12 Months Post Implantation
Population: The primary endpoint was compared between subjects in the qualifying with elevated NT-proBNP/BNP levels only group and subjects in the qualifying with prior HF hospitalization only group, but excluding primary endpoint events adjudicated as either related or possibly related to COVID-19.
Measure: Number; unit: events per patient-year
Groups:
- Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID-19 Related Events]; Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID-19 Related or Possibly Related Events]: All subjects had prior elevated NT-proBNP/BNP only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm - Previous HF Hospitalization Only [Exclude COVID-19 Related Events]; Single Arm - Previous HF Hospitalization Only [Exclude COVID-19 Related or Possibly Related Events]: All subjects had prior HF hospitalization only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID-19 Related Events] | Single Arm - Previous HF Hospitalization Only [Exclude COVID-19 Related Events] | Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID-19 Related or Possibly Related Events] | Single Arm - Previous HF Hospitalization Only [Exclude COVID-19 Related or Possibly Related Events]
Number analyzed (Participants) | 452 | 549 | 452 | 549
events per patient-year | 0.381 | 0.746 | 0.377 | 0.737

9. Secondary Outcome: (Randomized Arm) Composite Outcome of (1) HFHs and (2) Intravenous Diuretic Visits
Description: The composite outcome of:
  1. The number of recurrent heart failure hospitalizations (HFHs)
  2. The number of emergency department/hospital outpatient observation visits (ED/OP) for intravenous diuretic therapy
  added together with equal weighting into a total number of events
Time Frame: 12 months post-implantation
Population: The secondary outcome (composite of HFH and ED/OP visits) was analyzed in the full cohort of endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 497 | 503
events per patient-year | 0.474 | 0.557
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group vs Randomized Arm - Control Group; Test type: Superiority; p = 0.0958, Anderson-Gill model (robust sandwich); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.70 to 1.03]

10. Secondary Outcome: (Randomized Arm) Composite Outcome of (1) HFHs and (2) Intravenous Diuretic Visits [Follow-up Based COVID-19 Sensitivity Analysis)
Description: as for outcome 9
Time Frame: as for outcome 2
Population: The secondary outcome (composite of HFH and ED/OP visits) limited to the follow-up period occurring prior to COVID-19 or during COVID-19 were analyzed in the full cohort of endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized. All subjects were assessed based on their follow-up time occurring pre- or during-COVID periods using a time-varying covariate. The Arm/Group Titles represent the follow-up time period.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group [Pre-COVID-19] | Randomized Arm - Control Group [Pre-COVID-19] | Randomized Arm - Treatment Group [During COVID-19] | Randomized Arm - Control Group [During COVID-19]
Number analyzed (Participants) | 497 | 503 | 497 | 503
events per patient-year | 0.450 | 0.595 | 0.539 | 0.455

11. Secondary Outcome: (Randomized Arm) Composite Outcome of (1) HFHs and (2) Intravenous Diuretic Visits [Subject Based COVID-19 Sensitivity Analysis)
Description: as for outcome 9
Time Frame: 12 Months Post Implantation
Population: The secondary outcome (composite of HFH and ED/OP visits) was analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group (Pre-COVID-19) | Randomized Arm - Control Group (Pre-COVID-19) | Randomized Arm - Treatment Group (During COVID-19) | Randomized Arm - Control Arm (During COVID-19)
Number analyzed (Participants) | 187 | 196 | 310 | 307
events per patient-year | 0.529 | 0.729 | 0.465 | 0.488

12. Secondary Outcome: (Randomized Arm) Composite Outcome of (1) HFHs and (2) Intravenous Diuretic Visits [Event Based COVID-19 Sensitivity Analysis)
Description: as for outcome 9
Time Frame: 12 Months Post Implantation
Population: The composite outcome was analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. All subjects were enrolled before COVID-19 period (March 13, 2020). The event based COVID-19 sensitivity analysis compares treatment effect by excluding events adjudicated as either related or possible related to COVID-19.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group [Excluding COVID-19 Related Events] | Randomized Arm - Control Group [Excluding COVID-19 Related Events] | Randomized Arm - Treatment Group [Excluding COVID-19 Related or Possibly Related Events] | Randomized Arm - Control Group [Excluding COVID-19 Related or Possibly Related Events]
Number analyzed (Participants) | 497 | 503 | 497 | 503
events per patient-year | 0.474 | 0.551 | 0.472 | 0.545

13. Secondary Outcome: (Randomized Arm) HFHs
Description: The number of recurrent HFHs
Time Frame: 12 months post-implantation
Population: The number of recurrent HFHs were analyzed within the full cohort of endpoint-contributing population, which includes subjects of NYHA class II/III/IV that were successfully implanted and randomized.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 497 | 503
events per patient-year | 0.410 | 0.497
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group vs Randomized Arm - Control Group; Test type: Superiority; p = 0.0644, Anderson-Gill model (robust sandwich); Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.68 to 1.01]

14. Secondary Outcome: (Randomized Arm) HFHs [Follow-up Based COVID-19 Sensitivity Analysis]
Description: The number of recurrent HFHs
Time Frame: as for outcome 2
Population: The number of recurrent HFHs limited to the follow-up period occurring prior to COVID-19 or during COVID-19 were analyzed within the full cohort of endpoint-contributing population, which includes subjects of NYHA class II/III/IV that were successfully implanted and randomized. All subjects were assessed based on their follow-up time occurring pre- or during-COVID periods using a time-varying covariate. The Arm/Group Titles represent the follow-up time period.
Measure: Number; unit: events per patient-year
Groups:
- Randomized Arm - Treatment Group [Pre-COVID]; Randomized Arm - Treatment Group [During COVID-19]: Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Randomized Arm - Control Group [Pre-COVID]; Randomized Arm - Control Group [During COVID-19]: Management of subjects per standard of care (signs, symptoms, weight etc.) without knowledge of PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Randomized Arm - Treatment Group [Pre-COVID] | Randomized Arm - Control Group [Pre-COVID] | Randomized Arm - Treatment Group [During COVID-19] | Randomized Arm - Control Group [During COVID-19]
Number analyzed (Participants) | 497 | 503 | 497 | 503
events per patient-year | 0.380 | 0.525 | 0.490 | 0.414

15. Secondary Outcome: (Randomized Arm) HFHs [Subject Based COVID-19 Sensitivity Analysis]
Description: The number of recurrent HFHs
Time Frame: 12 Months Post-Implantation
Population: The number of recurrent HFHs was analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group (Pre-COVID-19) | Randomized Arm - Control Group (Pre-COVID-19) | Randomized Arm - Treatment Group (During COVID-19) | Randomized Arm - Control Arm (During COVID-19)
Number analyzed (Participants) | 187 | 196 | 310 | 307
events per patient-year | 0.467 | 0.666 | 0.399 | 0.428

16. Secondary Outcome: (Randomized Arm) HFHs [Event Based COVID-19 Sensitivity Analysis]
Description: The number of recurrent HFHs
Time Frame: 12 Months Post Implantation
Population: The number of recurrent HFHs was analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. All subjects were enrolled before COVID-19 period (March 13, 2020). The event based COVID-19 sensitivity analysis compares treatment effect by excluding events adjudicated as either related or possible related to COVID-19.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group [Excluding COVID-19 Related Events] | Randomized Arm - Control Group [Excluding COVID-19 Related Events] | Randomized Arm - Treatment Group [Excluding COVID-19 Related or Possibly Related Events] | Randomized Arm - Control Group [Excluding COVID-19 Related or Possibly Related Events]
Number analyzed (Participants) | 497 | 503 | 497 | 503
events per patient-year | 0.411 | 0.490 | 0.409 | 0.484

17. Secondary Outcome: (Randomized Arm) Intravenous Diuretic Visits
Description: The number of emergency department/hospital outpatient observation visits for intravenous diuretic therapy
Time Frame: 12 months post-implantation
Population: The number of ED/OP visits were analyzed in the full cohort of endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 497 | 503
events per patient-year | 0.065 | 0.063
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group vs Randomized Arm - Control Group; Test type: Superiority; p = 0.8867, Anderson-Gill model (robust sandwich); Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.61 to 1.77]

18. Secondary Outcome: (Randomized Arm) Intravenous Diuretic Visits [Follow-up Based COVID-19 Sensitivity Analysis]
Description: The number of emergency department/hospital outpatient observation visits for intravenous diuretic therapy
Time Frame: as for outcome 2
Population: The number of ED/OP visits limited to the follow-up period occurring prior to and during COVID-19 were analyzed in the full cohort of endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized. All subjects were assessed based on their follow-up time occurring pre- or during-COVID periods using a time-varying covariate. The Arm/Group Titles represent the follow-up time period.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group [Pre-COVID] | Randomized Arm - Control Group [Pre-COVID] | Randomized Arm - Treatment Group [During COVID-19] | Randomized Arm - Control Group [During COVID-19]
Number analyzed (Participants) | 497 | 503 | 497 | 503
events per patient-year | 0.074 | 0.073 | 0.048 | 0.041

19. Secondary Outcome: (Randomized Arm) Intravenous Diuretic Visits [Subject Based COVID-19 Sensitivity Analysis]
Description: The number of emergency department/hospital outpatient observation visits for intravenous diuretic therapy
Time Frame: 12 Months Post Implantation
Population: The outcome was analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group (Pre-COVID-19) | Randomized Arm - Control Group (Pre-COVID-19) | Randomized Arm - Treatment Group (During COVID-19) | Randomized Arm - Control Arm (During COVID-19)
Number analyzed (Participants) | 187 | 196 | 310 | 307
events per patient-year | 0.067 | 0.071 | 0.067 | 0.060

20. Secondary Outcome: (Randomized Arm) Intravenous Diuretic Visits [Event Based COVID-19 Sensitivity Analysis]
Description: The number of emergency department/hospital outpatient observation visits for intravenous diuretic therapy
Time Frame: 12 Months Post-Implantation
Population: The outcome was analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. All subjects were enrolled before COVID-19 period (March 13, 2020). The event based COVID-19 sensitivity analysis compares treatment effect by excluding events adjudicated as either related or possible related to COVID-19.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group [Excluding COVID-19 Related Events] | Randomized Arm - Control Group [Excluding COVID-19 Related Events] | Randomized Arm - Treatment Group [Excluding COVID-19 Related or Possibly Related Events] | Randomized Arm - Control Group [Excluding COVID-19 Related or Possibly Related Events]
Number analyzed (Participants) | 497 | 503 | 497 | 503
events per patient-year | 0.065 | 0.063 | 0.065 | 0.063

21. Secondary Outcome: (Randomized Arm) All-cause Mortality
Description: The number of deaths of any cause
Time Frame: 12 months post-implantation
Population: The number of death events of any cause were analyzed in the full cohort of endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 497 | 503
events per patient-year | 0.094 | 0.086
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group vs Randomized Arm - Control Group; Test type: Superiority; p = 0.7119, Anderson-Gill model (robust sandwich); Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.70 to 1.70]

22. Secondary Outcome: (Randomized Arm) All-cause Mortality [Follow-up Based COVID-19 Sensitivity Analysis]
Description: The number of deaths of any cause
Time Frame: as for outcome 2
Population: The number of death events of any cause limited to the follow-up period occurring prior to and during COVID-19 were analyzed in the full cohort of endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized. All subjects were assessed based on their follow-up time occurring pre- or during-COVID periods using a time-varying covariate. The Arm/Group Titles represent the follow-up time period.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group [Pre-COVID] | Randomized Arm - Control Group [Pre-COVID] | Randomized Arm - Treatment Group [During COVID-19] | Randomized Arm - Control Group [During COVID-19]
Number analyzed (Participants) | 497 | 503 | 497 | 503
events per patient-year | 0.110 | 0.088 | 0.067 | 0.085

23. Secondary Outcome: (Randomized Arm) All-cause Mortality [Subject Based COVID-19 Sensitivity Analysis]
Description: The number of deaths of any cause
Time Frame: 12 Months Post-Implantation
Population: The mortality events were analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group (Pre-COVID-19) | Randomized Arm - Control Group (Pre-COVID-19) | Randomized Arm - Treatment Group (During COVID-19) | Randomized Arm - Control Arm (During COVID-19)
Number analyzed (Participants) | 187 | 196 | 310 | 307
events per patient-year | 0.200 | 0.161 | 0.044 | 0.053

24. Secondary Outcome: (Randomized Arm) All-cause Mortality [Event Based COVID-19 Sensitivity Analysis]
Description: The number of deaths of any cause
Time Frame: 12 Months Post-Implantation
Population: The mortality events were analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. All subjects were enrolled before COVID-19 period (March 13, 2020). The event based COVID-19 sensitivity analysis compares treatment effect by excluding events adjudicated as either related or possible related to COVID-19.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group [Excluding COVID-19 Related Events] | Randomized Arm - Control Group [Excluding COVID-19 Related Events] | Randomized Arm - Treatment Group [Excluding COVID-19 Related or Possibly Related Events] | Randomized Arm - Control Group [Excluding COVID-19 Related or Possibly Related Events]
Number analyzed (Participants) | 497 | 503 | 497 | 503
events per patient-year | 0.094 | 0.086 | 0.090 | 0.079

25. Secondary Outcome: (Randomized Arm) KCCQ-12
Description: Health status as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ-12)
  The Kansas City Cardiomyopathy Questionnaire (KCCQ-12) is a validated health-related quality of life measure for heart failure and was qualified by the FDA as a medical device development tool in 2017. The KCCQ-12 quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life over a scale from 0 to 100. An overall summary score (OSS) is derived by averaging scores from each domain, with a higher score reflecting a better health status.
  Change from baseline KCCQ-12 scores were evaluated at 6 and 12-month visits.
Time Frame: Baseline, 6, and 12 months post-implantation
Population: Subjects that have a baseline value and at least one value at either 6- or 12-month visits were analyzed. The Least Square Means (LSM) difference in KCCQ-12 Overall Summary Score at 6 months, and 12 months visits from baseline during overall follow-up in Treatment and Control groups were analyzed using a mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Randomized Arm - Treatment Group (6 Month); Randomized Arm - Treatment Group (12 Month): Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Randomized Arm - Control Group (6 Month); Randomized Arm - Control Group (12 Month): Management of subjects per standard of care (signs, symptoms, weight etc.) without knowledge of PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Randomized Arm - Treatment Group (6 Month) | Randomized Arm - Control Group (6 Month) | Randomized Arm - Treatment Group (12 Month) | Randomized Arm - Control Group (12 Month)
Number analyzed (Participants) | 458 | 455 | 458 | 455
scores on a scale | 7.36 (1.01) | 6.01 (1.02) | 4.77 (1.03) | 4.14 (1.05)
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group (6 Month) vs Randomized Arm - Control Group (6 Month); Test type: Superiority; p = 0.3484, t-test, 1 sided; Mean Difference (Final Values) = -1.35, 95% CI 2-sided [-4.16 to 1.47], Standard Error of Mean 1.44
Statistical Analysis 2: Comparison: Randomized Arm - Treatment Group (12 Month) vs Randomized Arm - Control Group (12 Month); Test type: Superiority; p = 0.6684, t-test, 1 sided; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-3.51 to 2.26], Standard Error of Mean 1.47

26. Secondary Outcome: (Randomized Arm) KCCQ-12 (Subject Based COVID-19 Sensitivity Analysis)
Description: Health status as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) The Kansas City Cardiomyopathy Questionnaire (KCCQ-12) is a validated health-related quality of life measure for heart failure and was qualified by the FDA as a medical device development tool in 2017. The KCCQ-12 quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life over a scale from 0 to 100. An overall summary score (OSS) is derived by averaging scores from each domain, with a higher score reflecting a better health status.
  Descriptive statistics of KCCQ-12 scores at baseline, 6 and 12-month visits were reported.
Time Frame: Baseline, 6, and 12 months post-implantation
Population: The KCCQ-12 score at baseline, 6 months, and 12 months were analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Randomized Arm - Treatment Group (Baseline) [Pre-COVID-19]; Randomized Arm - Treatment Group (6 Month) [Pre-COVID-19]; Randomized Arm - Treatment Group (12 Month) [Pre-COVID-19]: Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending prior to COVID-19.
- Randomized Arm - Control Group (Baseline) [Pre-COVID-19]; Randomized Arm - Control Group (6 Month) [Pre-COVID-19]; Randomized Arm - Control Group (12 Month) [Pre-COVID-19]: Management of subjects per standard of care (signs, symptoms, weight etc.) without knowledge of PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending prior to COVID-19.
- Randomized Arm - Treatment Group (Baseline) [During COVID-19]; Randomized Arm - Treatment Group (6 Month) [During COVID-19]; Randomized Arm - Treatment Group (12 Month) [During COVID-19]: Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending during COVID-19.
- Randomized Arm - Control Group (Baseline) [During COVID-19]; Randomized Arm - Control Group (6 Month) [During COVID-19]; Randomized Arm - Control Group (12 Month) [During COVID-19]: Management of subjects per standard of care (signs, symptoms, weight etc.) without knowledge of PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending during COVID-19.
Arm/Group | Randomized Arm - Treatment Group (Baseline) [Pre-COVID-19] | Randomized Arm - Control Group (Baseline) [Pre-COVID-19] | Randomized Arm - Treatment Group (6 Month) [Pre-COVID-19] | Randomized Arm - Control Group (6 Month) [Pre-COVID-19] | Randomized Arm - Treatment Group (12 Month) [Pre-COVID-19] | Randomized Arm - Control Group (12 Month) [Pre-COVID-19] | Randomized Arm - Treatment Group (Baseline) [During COVID-19] | Randomized Arm - Control Group (Baseline) [During COVID-19] | Randomized Arm - Treatment Group (6 Month) [During COVID-19] | Randomized Arm - Control Group (6 Month) [During COVID-19] | Randomized Arm - Treatment Group (12 Month) [During COVID-19] | Randomized Arm - Control Group (12 Month) [During COVID-19]
Number analyzed (Participants) | 187 | 192 | 154 | 156 | 140 | 140 | 307 | 305 | 297 | 287 | 283 | 271
scores on a scale | 54.8 (25.4) | 56.4 (23.9) | 65.1 (24.3) | 63.6 (24.6) | 62.0 (24.0) | 62.9 (22.2) | 55.0 (23.6) | 53.9 (23.6) | 62.5 (24.3) | 60.3 (24.7) | 61.3 (24.7) | 58.2 (24.7)

27. Secondary Outcome: (Randomized Arm) EQ-5D-5L
Description: Health status as assessed by the EuroQol 5-Dimension, 5-Level (EQ-5D-5L) Questionnaire
  The EQ-5D-5L Questionnaire is a standardized measure of health status that consists of a descriptive system and a visual analog score (VAS). The VAS records the subject's self-rated health status which ranges from a score of 0 (worst health you can imagine) to 100 (best health you can imagine). A higher VAS score represents a better quality of life.
Time Frame: Baseline, 6, and 12 months post-implantation
Population: Subjects that have a baseline value and at least one value at either 6- or 12-month visits were analyzed. The Least Square Means (LSM) difference in EQ-5D-5L VAS at 6 months and 12 months visits from baseline during overall follow-up for Treatment and Control groups were analyzed using a mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Randomized Arm - Treatment Group (6 Month) | Randomized Arm - Control Group (6 Month) | Randomized Arm - Treatment Group (12 Month) | Randomized Arm - Control Group (12 Month)
Number analyzed (Participants) | 458 | 455 | 458 | 455
scores on a scale | 3.18 (0.97) | 3.20 (0.97) | 1.02 (0.99) | 2.50 (1.00)
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group (6 Month) vs Randomized Arm - Control Group (6 Month); Test type: Superiority; p = 0.9901, t-test, 1 sided; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-2.68 to 2.71], Standard Error of Mean 1.37
Statistical Analysis 2: Comparison: Randomized Arm - Treatment Group (12 Month) vs Randomized Arm - Control Group (12 Month); Test type: Superiority; p = 0.2947, t-test, 1 sided; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [-1.29 to 4.24], Standard Error of Mean 1.41

28. Secondary Outcome: (Randomized Arm) EQ-5D-5L (Subject Based COVID-19 Sensitivity Analysis)
Description: as for outcome 27
Time Frame: Baseline, 6, and 12 months post-implantation
Population: The EQ-5D-5L score at baseline, 6 months, and 12 months were analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Randomized Arm - Treatment Group (Baseline) [Pre-COVID-19] | Randomized Arm - Control Group (Baseline) [Pre-COVID-19] | Randomized Arm - Treatment Group (6 Month) [Pre-COVID-19] | Randomized Arm - Control Group (6 Month) [Pre-COVID-19] | Randomized Arm - Treatment Group (12 Month) [Pre-COVID-19] | Randomized Arm - Control Group (12 Month) [Pre-COVID-19] | Randomized Arm - Treatment Group (Baseline) [During COVID-19] | Randomized Arm - Control Group (Baseline) [During COVID-19] | Randomized Arm - Treatment Group (6 Month) [During COVID-19] | Randomized Arm - Control Group (6 Month) [During COVID-19] | Randomized Arm - Treatment Group (12 Month) [During COVID-19] | Randomized Arm - Control Group (12 Month) [During COVID-19]
Number analyzed (Participants) | 187 | 192 | 154 | 156 | 140 | 141 | 308 | 305 | 297 | 288 | 283 | 271
scores on a scale | 66.5 (20.3) | 67.3 (18.9) | 71.7 (18.3) | 71.2 (20.0) | 68.3 (20.9) | 71.5 (18.5) | 66.2 (18.1) | 63.4 (19.7) | 69.5 (19.2) | 67.1 (20.6) | 68.8 (19.8) | 66.4 (21.9)

29. Secondary Outcome: (Randomized Arm) 6MHW Test
Description: Six Minute Hall Walk (6MHW) Test Distance
Time Frame: Baseline, 6, and 12 months post-implantation
Population: Subjects that have a baseline value and at least one value at either 6- or 12-month visits were analyzed. Subjects who were unable to walk due to heart failure symptoms were assigned zero meters. The Least Square Means (LSM) difference in 6MHW distance at 6 months and 12 months from baseline in both Treatment and Control groups during the overall follow-up period were analyzed using a mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: meters, m
Arm/Group | Randomized Arm - Treatment Group (6 Month) | Randomized Arm - Control Group (6 Month) | Randomized Arm - Treatment Group (12 Month) | Randomized Arm - Control Group (12 Month)
Number analyzed (Participants) | 382 | 397 | 382 | 397
meters, m | -1.13 (5.25) | 3.01 (5.16) | -13.02 (5.54) | -10.09 (5.50)
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group (6 Month) vs Randomized Arm - Control Group (6 Month); Test type: Superiority; p = 0.5741, t-test, 1 sided; Mean Difference (Final Values) = 4.14, 95% CI 2-sided [-10.32 to 18.60], Standard Error of Mean 7.36
Statistical Analysis 2: Comparison: Randomized Arm - Treatment Group (12 Month) vs Randomized Arm - Control Group (12 Month); Test type: Superiority; p = 0.7077, t-test, 1 sided; Mean Difference (Final Values) = 2.93, 95% CI 2-sided [-12.41 to 18.27], Standard Error of Mean 7.81

30. Secondary Outcome: (Randomized Arm) 6MHW Test (Subject Based COVID-19 Sensitivity Analysis)
Description: Six Minute Hall Walk (6MHW) Test Distance
Time Frame: Baseline, 6, and 12 months post-implantation
Population: The 6MHW distance at baseline, 6 months, and 12 months were analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV that were successfully implanted and randomized into Treatment or Control groups. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: meters, m
Arm/Group | Randomized Arm - Treatment Group (Baseline) [Pre-COVID-19] | Randomized Arm - Control Group (Baseline) [Pre-COVID-19] | Randomized Arm - Treatment Group (6 Month) [Pre-COVID-19] | Randomized Arm - Control Group (6 Month) [Pre-COVID-19] | Randomized Arm - Treatment Group (12 Month) [Pre-COVID-19] | Randomized Arm - Control Group (12 Month) [Pre-COVID-19] | Randomized Arm - Treatment Group (Baseline) [During COVID-19] | Randomized Arm - Control Group (Baseline) [During COVID-19] | Randomized Arm - Treatment Group (6 Month) [During COVID-19] | Randomized Arm - Control Group (6 Month) [During COVID-19] | Randomized Arm - Treatment Group (12 Month) [During COVID-19] | Randomized Arm - Control Group (12 Month) [During COVID-19]
Number analyzed (Participants) | 179 | 187 | 138 | 147 | 124 | 130 | 295 | 295 | 200 | 203 | 171 | 168
meters, m | 227 (117.8) | 243.8 (124.7) | 239.3 (123.5) | 260.8 (120.8) | 230.4 (133.2) | 245.1 (136.1) | 240.2 (121.5) | 220.6 (121.3) | 249.8 (129.1) | 244.7 (135.6) | 246.0 (130.0) | 230.7 (135.3)

31. Secondary Outcome: (Randomized Arm) Safety: Freedom From DSRCs
Description: Freedom from device/system related complications (DSRCs)
Time Frame: 12 months post-implantation
Population: The overall freedom from DSRCs across the endpoint-contributing population were analyzed. The analysis population included all subjects in the efficacy population of the Randomized Arm (i.e. Randomized to Treatment and Control group).
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 497 | 503
Participants | 494 | 498

32. Secondary Outcome: (Single Arm) Composite Outcome of (1) HFHs and (2) Intravenous Diuretic Visits
Description: The composite outcome of:
  1. The number of recurrent HFHs
  2. The number of emergency department/hospital outpatient observation visits for intravenous diuretic therapy
  added together with equal weighting into a total number of events
Time Frame: 12 months post-implantation
Population: The secondary endpoint was compared between subjects qualifying with elevated NT-proBNP/BNP levels only and subjects qualifying with a prior HF hospitalization only.
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only
Number analyzed (Participants) | 452 | 549
events per patient-year | 0.288 | 0.630
Statistical Analysis 1: Comparison: Single Arm - Elevated NT-proBNP/BNP Only vs Single Arm - Previous HF Hospitalization Only; Test type: Equivalence — Clinical equivalence was met if the lower limit of the CI of ln(HR) for the primary endpoint in Elevated NT-proBNP/BNP only vs. prior HFH only subjects is > -0.2877 and the upper limit is < 0.2877; Hazard Ratio (HR) = 0.46, 90% CI 2-sided [0.38 to 0.55]

33. Secondary Outcome: (Single Arm) Composite Outcome of (1) HFHs and (2) Intravenous Diuretic Visits [Follow-up Based COVID-19 Sensitivity Analysis]
Description: as for outcome 32
Time Frame: as for outcome 6
Population: The secondary outcome events limited to the follow-up period were compared between subjects in the qualifying with elevated NT-proBNP/BNP levels only group and subjects in the qualifying with prior HF hospitalization only group. Subjects were assessed based on their follow-up time occurring pre- or during-COVID periods using a time-varying covariate. The Arm/Group Titles represent the follow-up time period.
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Prior to COVID-19] | Single Arm - Previous HF Hospitalization Only [Prior to COVID-19] | Single Arm - Elevated NT-proBNP/BNP Only [During COVID-19] | Single Arm - Previous HF Hospitalization Only [During COVID-19]
Number analyzed (Participants) | 452 | 549 | 452 | 549
events per patient-year | 0.211 | 0.677 | 0.303 | 0.616

34. Secondary Outcome: (Single Arm) Composite Outcome of (1) HFHs and (2) Intravenous Diuretic Visits [Subject Based COVID-19 Sensitivity Analysis]
Description: as for outcome 32
Time Frame: 12 Months Post Implantation
Population: The results were compared between subjects in the qualifying with elevated NT-proBNP/BNP levels only group and subjects in the qualifying with prior HF hospitalization only group. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only (Pre-COVID-19) | Single Arm - Previous HF Hospitalization Only (Pre-COVID-19) | Single Arm - Elevated NT-proBNP/BNP Only (During COVID-19) | Single Arm - Previous HF Hospitalization Only (During COVID-19)
Number analyzed (Participants) | 25 | 69 | 427 | 480
events per patient-year | 0.436 | 1.520 | 0.286 | 0.583

35. Secondary Outcome: (Single Arm) Composite Outcome of (1) HFHs and (2) Intravenous Diuretic Visits [Event Based COVID-19 Sensitivity Analysis]
Description: as for outcome 32
Time Frame: 12 Months Post Implantation
Population: The results were compared between subjects in the qualifying with elevated NT-proBNP/BNP levels only group and subjects in the qualifying with prior HF hospitalization only group, but excluding primary endpoint events adjudicated as either related or possibly related to COVID-19.
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID-19 Related Events] | Single Arm - Previous HF Hospitalization Only [Exclude COVID-19 Related Events] | Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID-19 Related or Possibly Related Events] | Single Arm - Previous HF Hospitalization Only [Exclude COVID-19 Related or Possibly Related Events]
Number analyzed (Participants) | 452 | 549 | 452 | 549
events per patient-year | 0.282 | 0.624 | 0.277 | 0.617

36. Secondary Outcome: (Single Arm) Intravenous Diuretic Visits
Description: The number of emergency department/hospital outpatient observation (ED/OP) visits for intravenous diuretic therapy
Time Frame: 12 months post-implantation
Population: The secondary endpoint was analyzed in the endpoint-contributing populations, which consists of subjects with successful implantation in three qualifying groups: elevated NT-proBNP/BNP only, previous HF hospitalization only or both elevated NT-proBNP/BNP and previous HF hospitalization. Annualized event rate was estimated from the Andersen-Gill model.
Measure: Number; unit: events per patient-year
Groups:
- Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization: All subjects had prior elevated NT-proBNP/BNP and HF hospitalization with successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 549 | 343
events per patient-year | 0.027 | 0.077 | 0.123
Statistical Analysis 1: Comparison: Single Arm - Elevated NT-proBNP/BNP Only vs Single Arm - Previous HF Hospitalization Only vs Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization; Test type: Other; p < 0.0001, ANOVA

37. Secondary Outcome: (Single Arm) Intravenous Diuretic Visits [Follow-up Based COVID-19 Sensitivity Analysis]
Description: The number of emergency department/hospital outpatient observation (ED/OP) visits for intravenous diuretic therapy
Time Frame: as for outcome 6
Population: The endpoints limited to the follow-up period was analyzed in the endpoint-contributing populations, which consists of subjects with successful implantation in three qualifying groups: elevated NT-proBNP/BNP only, previous HF hospitalization only or both elevated NT-proBNP/BNP and previous HF hospitalization. Subjects were assessed based on their follow-up time occurring pre- or during-COVID periods using a time-varying covariate. The Arm/Group Titles represent the follow-up time period.
Measure: Number; unit: events per patient-year
Groups:
- Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Prior to COVID-19]; Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [During COVID-19]: All subjects had prior elevated NT-proBNP/BNP and HF hospitalization with successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Prior to COVID-19] | Single Arm - Previous HF Hospitalization Only [Prior to COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Prior to COVID-19] | Single Arm - Elevated NT-proBNP/BNP Only [During COVID-19] | Single Arm - Previous HF Hospitalization Only [During COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [During COVID-19]
Number analyzed (Participants) | 452 | 549 | 343 | 452 | 549 | 343
events per patient-year | 0.055 | 0.064 | 0.199 | 0.024 | 0.088 | 0.114

38. Secondary Outcome: (Single Arm) Intravenous Diuretic Visits [Subject Based COVID-19 Sensitivity Analysis]
Description: The number of emergency department/hospital outpatient observation (ED/OP) visits for intravenous diuretic therapy
Time Frame: 12 months post-implantation
Population: The event was compared between subjects in the three qualifying groups: elevated NT-proBNP/BNP only, previous HF hospitalization only or both elevated NT-proBNP/BNP and previous HF hospitalization. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Number; unit: events per patient-year
Groups:
- Single Arm - Elevated NT-proBNP/BNP Only [Pre-COVID-19]: All subjects had prior elevated NT-proBNP/BNP only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending prior to COVID-19.
- Single Arm - Previous HF Hospitalization Only [Pre-COVID-19]: All subjects had prior HF hospitalization only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending prior to COVID-19.
- Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Pre-COVID-19]: All subjects had prior elevated NT-proBNP/BNP and HF hospitalization with successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending prior to COVID-19.
- Single Arm - Elevated NT-proBNP/BNP Only [During COVID-19]: All subjects had prior elevated NT-proBNP/BNP only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending during COVID-19.
- Single Arm - Previous HF Hospitalization Only [During COVID-19]: All subjects had prior HF hospitalization only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending during COVID-19.
- Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [During COVID-19]: All subjects had prior elevated NT-proBNP/BNP and HF hospitalization with successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Subjects with follow-up ending during COVID-19.
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Pre-COVID-19] | Single Arm - Previous HF Hospitalization Only [Pre-COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Pre-COVID-19] | Single Arm - Elevated NT-proBNP/BNP Only [During COVID-19] | Single Arm - Previous HF Hospitalization Only [During COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [During COVID-19]
Number analyzed (Participants) | 25 | 69 | 50 | 427 | 480 | 293
events per patient-year | 0.213 | 0.082 | 0.422 | 0.021 | 0.080 | 0.101

39. Secondary Outcome: (Single Arm) Intravenous Diuretic Visits [Event Based COVID-19 Sensitivity Analysis]
Description: The number of emergency department/hospital outpatient observation (ED/OP) visits for intravenous diuretic therapy
Time Frame: 12 Months Post Implantation
Population: The event was compared between subjects in the three qualifying groups: elevated NT-proBNP/BNP only, previous HF hospitalization only or both elevated NT-proBNP/BNP and previous HF hospitalization, but excluding events adjudicated as either related or possibly related to COVID-19.
Measure: Number; unit: events per patient-year
Groups:
- Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID Related Events]; Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID Related/Possibly Related Events]: All subjects had prior elevated NT-proBNP/BNP only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm - Previous HF Hospitalization Only [Exclude COVID Related Events]; Single Arm - Previous HF Hospitalization Only [Exclude COVID Related/Possibly Related Events]: All subjects had prior HF hospitalization only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Exclude COVID Related Events]; Single Arm - Elevated NT-proBNP/BNP and Previous HFH [Exclude COVID Related/Possibly Related Events]: All subjects had prior elevated NT-proBNP/BNP and HF hospitalization with successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID Related Events] | Single Arm - Previous HF Hospitalization Only [Exclude COVID Related Events] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Exclude COVID Related Events] | Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID Related/Possibly Related Events] | Single Arm - Previous HF Hospitalization Only [Exclude COVID Related/Possibly Related Events] | Single Arm - Elevated NT-proBNP/BNP and Previous HFH [Exclude COVID Related/Possibly Related Events]
Number analyzed (Participants) | 452 | 549 | 343 | 452 | 549 | 343
events per patient-year | 0.027 | 0.077 | 0.123 | 0.027 | 0.075 | 0.119

40. Secondary Outcome: (Single Arm) HFHs
Description: The number of HFHs
Time Frame: 12 months post-implantation
Population: as for outcome 36
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 549 | 343
events per patient-year | 0.263 | 0.557 | 0.797
Statistical Analysis 1: Comparison: Single Arm - Elevated NT-proBNP/BNP Only vs Single Arm - Previous HF Hospitalization Only vs Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization; Test type: Other; p < 0.0001, ANOVA

41. Secondary Outcome: (Single Arm) HFHs [Follow-Up Based COVID-19 Sensitivity Analysis]
Description: The number of heart failure hospitalizations (HFHs)
Time Frame: as for outcome 6
Population: The secondary outcome events limited to the follow-up period occurring prior to COVID-19 or during COVID-19 was compared between subjects in the three qualifying groups: elevated NT-proBNP/BNP only, previous HF hospitalization only or both elevated NT-proBNP/BNP and previous HF hospitalization. Subjects were assessed based on their follow-up time occurring pre- or during-COVID periods using a time-varying covariate. The Arm/Group Titles represent the follow-up time period.
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Prior to COVID-19] | Single Arm - Previous HF Hospitalization Only [Prior to COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Prior to COVID-19] | Single Arm - Elevated NT-proBNP/BNP Only [During COVID-19] | Single Arm - Previous HF Hospitalization Only [During COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [During COVID-19]
Number analyzed (Participants) | 452 | 549 | 343 | 452 | 549 | 343
events per patient-year | 0.214 | 0.804 | 1.211 | 0.280 | 0.529 | 0.732

42. Secondary Outcome: (Single Arm) HFHs [Subject Based COVID-19 Sensitivity Analysis]
Description: The number of heart failure hospitalizations (HFHs)
Time Frame: 12 Months Post Implantation
Population: The HFH event was compared between subjects in the three qualifying groups: elevated NT-proBNP/BNP only, previous HF hospitalization only or both elevated NT-proBNP/BNP and previous HF hospitalization. The "Pre-COVID-19" Arms/Groups assess participants that completed study participation prior to the start of the COVID-19 pandemic, and the "During COVID-19" Arms/Groups assess participants that completed study participation during the COVID-19 pandemic.
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Pre-COVID-19] | Single Arm - Previous HF Hospitalization Only [Pre-COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Pre-COVID-19] | Single Arm - Elevated NT-proBNP/BNP Only [During COVID-19] | Single Arm - Previous HF Hospitalization Only [During COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [During COVID-19]
Number analyzed (Participants) | 25 | 69 | 50 | 427 | 480 | 293
events per patient-year | 0.175 | 1.132 | 1.660 | 0.269 | 0.510 | 0.719

43. Secondary Outcome: (Single Arm) HFHs [Event Based COVID-19 Sensitivity Analysis]
Description: The number of heart failure hospitalizations (HFHs)
Time Frame: 12 Months Post Implantation
Population: The HFH event was compared between subjects in the three qualifying groups: elevated NT-proBNP/BNP only, previous HF hospitalization only or both elevated NT-proBNP/BNP and previous HF hospitalization, but excluding events adjudicated as either related or possibly related to COVID-19.
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID Related Events] | Single Arm - Previous HF Hospitalization Only [Exclude COVID Related Events] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Exclude COVID Related Events] | Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID Related/Possibly Related Events] | Single Arm - Previous HF Hospitalization Only [Exclude COVID Related/Possibly Related Events] | Single Arm - Elevated NT-proBNP/BNP and Previous HFH [Exclude COVID Related/Possibly Related Events]
Number analyzed (Participants) | 452 | 549 | 343 | 452 | 549 | 343
events per patient-year | 0.257 | 0.552 | 0.790 | 0.252 | 0.545 | 0.749

44. Secondary Outcome: (Single Arm) All-cause Mortality
Description: The number of deaths of any cause
Time Frame: 12 months post-implantation
Population: as for outcome 36
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 549 | 343
events per patient-year | 0.113 | 0.146 | 0.243
Statistical Analysis 1: Comparison: Single Arm - Elevated NT-proBNP/BNP Only vs Single Arm - Previous HF Hospitalization Only vs Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization; Test type: Other; p = 0.0001, ANOVA

45. Secondary Outcome: (Single Arm) All-cause Mortality [Follow-Up Based COVID-19 Sensitivity Analysis]
Description: The number of deaths of any cause
Time Frame: as for outcome 6
Population: The event limited to the follow-up period occurring prior to COVID-19 or during COVID-19 was compared between subjects in the three qualifying groups: elevated NT-proBNP/BNP only, previous HF hospitalization only or both elevated NT-proBNP/BNP and previous HF hospitalization. Subjects were assessed based on their follow-up time occurring pre- or during-COVID periods using a time-varying covariate. The Arm/Group Titles represent the follow-up time period.
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Prior to COVID-19] | Single Arm - Previous HF Hospitalization Only [Prior to COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Prior to COVID-19] | Single Arm - Elevated NT-proBNP/BNP Only [During COVID-19] | Single Arm - Previous HF Hospitalization Only [During COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [During COVID-19]
Number analyzed (Participants) | 452 | 549 | 343 | 452 | 549 | 343
events per patient-year | 0.050 | 0.182 | 0.272 | 0.123 | 0.135 | 0.233

46. Secondary Outcome: (Single Arm) All-cause Mortality [Subject Based COVID-19 Sensitivity Analysis]
Description: The number of deaths of any cause
Time Frame: 12 Months Post Implantation
Population: as for outcome 42
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Pre-COVID-19] | Single Arm - Previous HF Hospitalization Only [Pre-COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Pre-COVID-19] | Single Arm - Elevated NT-proBNP/BNP Only [During COVID-19] | Single Arm - Previous HF Hospitalization Only [During COVID-19] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [During COVID-19]
Number analyzed (Participants) | 25 | 69 | 50 | 427 | 480 | 293
events per patient-year | 0.147 | 0.384 | 0.583 | 0.113 | 0.120 | 0.202

47. Secondary Outcome: (Single Arm) All-cause Mortality [Event Based COVID-19 Sensitivity Analysis]
Description: The number of deaths of any cause
Time Frame: 12 Months Post Implantation
Population: as for outcome 39
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID Related Events] | Single Arm - Previous HF Hospitalization Only [Exclude COVID Related Events] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [Exclude COVID Related Events] | Single Arm - Elevated NT-proBNP/BNP Only [Exclude COVID Related/Possibly Related Events] | Single Arm - Previous HF Hospitalization Only [Exclude COVID Related/Possibly Related Events] | Single Arm - Elevated NT-proBNP/BNP and Previous HFH [Exclude COVID Related/Possibly Related Events]
Number analyzed (Participants) | 452 | 549 | 343 | 452 | 549 | 343
events per patient-year | 0.105 | 0.125 | 0.231 | 0.105 | 0.123 | 0.227

48. Secondary Outcome: (Single Arm) Safety: Freedom From DSRCs
Description: Proportion of subjects with freedom from device/system related complications (DSRCs)
Time Frame: 12 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 549 | 343
Participants | 451 | 548 | 342

49. Secondary Outcome: (Single Arm) HFHs Post- vs. Pre-implantation [Elevated NT-proBNP/BNP Only Group]
Description: The number of HFHs at 12 months post-implantation compared to the number of HFHs in the 12 months prior to implantation
Time Frame: 12 months post-implantation vs 12 months pre-implantation
Population: All subjects met qualification criteria of prior elevated NT-proBNP/BNP only and had successful implantation of CardioMEMS™ HF System.
Measure: Number; unit: events per patient-year
Groups:
- Single Arm - Elevated NT-proBNP/BNP Only (One Year Prior to Implant); Single Arm - Elevated NT-proBNP/BNP (One Year After Implant): All subjects had prior elevated NT-proBNP/BNP only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only (One Year Prior to Implant) | Single Arm - Elevated NT-proBNP/BNP (One Year After Implant)
Number analyzed (Participants) | 452 | 452
events per patient-year | 0 | 0.265

50. Secondary Outcome: (Single Arm) HFHs Post- vs. Pre-implantation [Previous HF Hospitalization Only Group]
Description: The number of HFHs at 12 months post-implantation compared to the number of HFHs in the 12 months prior to implantation
Time Frame: 12 months post-implantation vs 12 months pre-implantation
Population: All subjects met qualification criteria of previous HF hospitalization only and had successful implantation of CardioMEMS™ HF System.
Measure: Number; unit: events per patient-year
Groups:
- Single Arm - Previous HF Hospitalization Only (One Year Prior to Implant): All subjects had previous HF hospitalization only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm - Previous HF Hospitalization (One Year After Implant): All subjects had previous HF hospitalization and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Single Arm - Previous HF Hospitalization Only (One Year Prior to Implant) | Single Arm - Previous HF Hospitalization (One Year After Implant)
Number analyzed (Participants) | 549 | 549
events per patient-year | 1.170 | 0.540
Statistical Analysis 1: Comparison: Single Arm - Previous HF Hospitalization Only (One Year Prior to Implant) vs Single Arm - Previous HF Hospitalization (One Year After Implant); Test type: Other; p < 0.0001, Anderson-Gill model (robust sandwich); Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.39 to 0.54]

51. Secondary Outcome: (Single Arm) HFHs Post- vs. Pre-implantation [Elevated NT-proBNP/BNP and Previous HF Hospitalization Group]
Description: The number of HFHs at 12 months post-implantation compared to the number of HFHs in the 12 months prior to implantation
Time Frame: 12 months post-implantation vs 12 months pre-implantation
Population: All subjects met qualification criteria of elevated NT-proBNP/BNP and previous HF hospitalization and had successful implantation of CardioMEMS™ HF System.
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Previous HF Hospitalization Only (One Year Prior to Implant) | Single Arm - Previous HF Hospitalization (One Year After Implant)
Number analyzed (Participants) | 343 | 343
events per patient-year | 1.380 | 0.874
Statistical Analysis 1: Comparison: Single Arm - Previous HF Hospitalization Only (One Year Prior to Implant) vs Single Arm - Previous HF Hospitalization (One Year After Implant); Test type: Other; p < 0.001, Anderson-Gill model (robust sandwich); Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.53 to 0.76]

52. Other Pre Specified Outcome: (Randomized Arm) Cardiovascular Mortality
Description: The number of deaths with cardiovascular cause
Time Frame: 12 months post-implantation
Population: The number of deaths that were cardiovascular in nature were analyzed in the endpoint contributing population, which includes subjects of NYHA class II/III/IV with successful implantation and randomized.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 497 | 503
events per patient-year | 0.071 | 0.057

53. Other Pre Specified Outcome: (Randomized Arm) All-cause Hospitalizations
Description: The number of hospitalizations of any cause
Time Frame: 12 months post-implantation
Population: The number of all-cause hospitalizations were analyzed in the endpoint-contributing population, which included subjects of NYHA class II/III/IV with successful implantation and randomized.
Measure: Number; unit: events per patient-year
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 497 | 503
events per patient-year | 0.918 | 0.973

54. Other Pre Specified Outcome: (Randomized Arm) Frequency of Subject PA Pressure Uploads
Description: The frequency of subject uploads of PA pressure
Time Frame: 12 months post-implantation
Population: Subjects with at least one eligible day during the analysis period are included in the analysis. The daily compliance (percentage of eligible days in which a subject had a reading) and weekly compliance (percentage of weeks in which a subject had at least one reading) per subject were analyzed in the endpoint contributing population that had at least one reading post-discharge from the implantation. Days when subjects did not have any reading taken during the eligible days are counted as zeroes.
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 497 | 502
Percentage
  Daily compliance | 80.7 (20.4) | 73.8 (27.0)
  Weekly compliance | 95.1 (13.7) | 89.1 (21.7)

55. Other Pre Specified Outcome: (Randomized Arm) HF Medication Changes
Description: The number of changes in HF medications
Time Frame: 12 months post-implantation
Population: Within the endpoint-contributing population, which included subjects of NYHA class II/II/IV with successful implantation and randomized into Treatment and Control group, the number of subjects with medication changes and the number of medications changes were recorded by different classes of HF medications.
Measure: Number; unit: Number of medication changes
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 497 | 503
Number of medication changes
  Angiotensin-Converting Enzyme (ACE) Inhibitors: number analyzed (Participants) | 51 | 44
  Angiotensin-Converting Enzyme (ACE) Inhibitors | 109 | 76
  Angiotensin Receptor Blocker (ARB): number analyzed (Participants) | 55 | 45
  Angiotensin Receptor Blocker (ARB) | 94 | 80
  Angiotensin Receptor-Neprilysin Inhibitor (ARNi): number analyzed (Participants) | 78 | 63
  Angiotensin Receptor-Neprilysin Inhibitor (ARNi) | 194 | 120
  Beta Blockers: number analyzed (Participants) | 162 | 156
  Beta Blockers | 370 | 339
  Aldosterone Antagonists: number analyzed (Participants) | 130 | 101
  Aldosterone Antagonists | 323 | 190
  Diuretics: number analyzed (Participants) | 431 | 328
  Diuretics | 3961 | 2064
  Nitrates: number analyzed (Participants) | 65 | 53
  Nitrates | 169 | 101
  Vasodilators: number analyzed (Participants) | 64 | 50
  Vasodilators | 146 | 83
  SGLT2 Inhibitor: number analyzed (Participants) | 9 | 5
  SGLT2 Inhibitor | 9 | 6
  Calcium Channel Blockers: number analyzed (Participants) | 48 | 36
  Calcium Channel Blockers | 77 | 65
  Digoxin: number analyzed (Participants) | 17 | 20
  Digoxin | 24 | 36
  Sinus Node If Channel Inhibitors: number analyzed (Participants) | 8 | 3
  Sinus Node If Channel Inhibitors | 12 | 4

56. Other Pre Specified Outcome: (Randomized Arm) PA Pressure Measurements [Mixed Model Analysis]
Description: Changes in PA pressure relative to baseline for systolic, diastolic, and mean PA pressures analyzed using a mixed linear model at fixed time points (Baseline, 6 months, and 12 months) producing least-squares means.
Time Frame: Baseline through 12 months post-implantation
Population: Subjects that have a baseline value and at least one value at either 6- or 12-month visits were analyzed. The Least Square Means (LSM) difference in PA pressure measurements at 6 months and 12 months from baseline in both Treatment and Control groups during the overall follow-up period were analyzed using a mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Randomized Arm - Treatment Group (6 Month) | Randomized Arm - Control Group (6 Month) | Randomized Arm - Treatment Group (12 Month) | Randomized Arm - Control Group (12 Month)
Number analyzed (Participants) | 455 | 432 | 455 | 432
mmHg
  PA Systolic Pressure | -3.41 (0.44) | -1.87 (0.46) | -3.33 (0.46) | -2.70 (0.47)
  PA Diastolic pressure | -2.52 (0.27) | -1.73 (0.28) | -2.49 (0.28) | -2.29 (0.29)
  PA Mean Pressure | -2.90 (0.34) | -1.77 (0.35) | -2.80 (0.35) | -2.40 (0.36)
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group (6 Month) vs Randomized Arm - Control Group (6 Month); Comparisons of PA Systolic Pressure at 6 months between Treatment vs Control group; Test type: Superiority; p = 0.0160, Mixed Models Analysis; Least Square Means Difference (T vs C) = 1.53, 95% CI 2-sided [0.29 to 2.78], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: Randomized Arm - Treatment Group (6 Month) vs Randomized Arm - Control Group (6 Month); Comparisons of PA Diastolic Pressure at 6 months between Treatment vs Control group; Test type: Superiority; p = 0.0427, Mixed Models Analysis; Least Square Means Difference (T vs C) = 0.79, 95% CI 2-sided [0.03 to 1.56], Standard Error of Mean 0.39
Statistical Analysis 3: Comparison: Randomized Arm - Treatment Group (6 Month) vs Randomized Arm - Control Group (6 Month); Comparisons of PA Mean Pressure at 6 months between Treatment vs Control group; Test type: Superiority; p = 0.0188, Mixed Models Analysis; Least Square Means Difference (T vs C) = 1.13, 95% CI 2-sided [0.19 to 2.08], Standard Error of Mean 0.48
Statistical Analysis 4: Comparison: Randomized Arm - Treatment Group (12 Month) vs Randomized Arm - Control Group (12 Month); Comparisons of PA Systolic Pressure at 12 months between Treatment vs Control group; Test type: Superiority; p = 0.3405, Mixed Models Analysis; Least Square Means Difference (T vs C) = 0.63, 95% CI 2-sided [-0.66 to 1.92], Standard Error of Mean 0.66
Statistical Analysis 5: Comparison: Randomized Arm - Treatment Group (12 Month) vs Randomized Arm - Control Group (12 Month); Comparisons of PA Diastolic Pressure at 12 months between Treatment vs Control group; Test type: Superiority; p = 0.6174, Mixed Models Analysis; Least Square Means Difference (T vs C) = 0.20, 95% CI 2-sided [-0.59 to 0.99], Standard Error of Mean 0.40
Statistical Analysis 6: Comparison: Randomized Arm - Treatment Group (12 Month) vs Randomized Arm - Control Group (12 Month); Comparisons of PA Mean Pressure at 12 months between Treatment vs Control group; Test type: Superiority; p = 0.4231, Mixed Models Analysis; Least Square Means Difference (T vs C) = 0.40, 95% CI 2-sided [-0.58 to 1.38], Standard Error of Mean 0.50

57. Other Pre Specified Outcome: (Randomized Arm) PA Pressure Measurements [AUC Analysis]
Description: Changes in PA pressure relative to baseline for systolic, diastolic, and mean PA pressures analyzed using an area under the curve (AUC) analysis of change from baseline on all PA pressure readings through 12 months.
Time Frame: Baseline through 12 months post-implantation
Population: The PA pressure measurements were analyzed in the endpoint contributing population that had at least one reading post-discharge from the implantation.
Measure: Mean (Standard Deviation); unit: mmHg*Days
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 497 | 499
mmHg*Days
  PA Systolic Pressure | -945.0 (2328.9) | -621.2 (2242.3)
  PA Diastolic pressure | -690.5 (1405.1) | -566.1 (1360.6)
  PA Mean Pressure | -792.7 (1767.0) | -582.9 (1698.1)
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group vs Randomized Arm - Control Group; Comparison of PA Systolic Pressure AUC between Treatment and Control group; Test type: Superiority; p = 0.0214, t-test, 2 sided
Statistical Analysis 2: Comparison: Randomized Arm - Treatment Group vs Randomized Arm - Control Group; Comparison of PA Diastolic Pressure AUC between Treatment and Control group; Test type: Other; p = 0.1002, t-test, 2 sided
Statistical Analysis 3: Comparison: Randomized Arm - Treatment Group vs Randomized Arm - Control Group; Comparison of PA Mean Pressure AUC between Treatment and Control group; Test type: Other; p = 0.0402, t-test, 2 sided

58. Other Pre Specified Outcome: (Randomized Arm) BNP
Description: Change in BNP measurements from baseline
Time Frame: 6 months post-implantation
Population: Subjects that have a baseline value and at least one value at 6-month visit were analyzed. The Least Square Means (LSM) difference in BNP levels at 6 months from baseline in both Treatment and Control groups during the overall follow-up period were analyzed using a mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 235 | 221
pg/mL | -72.16 (52.46) | -34.96 (54.33)
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group vs Randomized Arm - Control Group; Comparisons of change from baseline in BNP levels at 6 months between Treatment vs Control group; Test type: Superiority; p = 0.6227, Mixed Models Analysis; Least Square Means Difference (T vs C) = 37.19, 95% CI 2-sided [-111.38 to 185.77], Standard Error of Mean 75.52

59. Other Pre Specified Outcome: (Randomized Arm) BNP
Description: Change in BNP measurements from baseline
Time Frame: 12 months post-implantation
Population: Subjects that have a baseline value and at least one value at 12-month visits were analyzed. The Least Square Means (LSM) difference in BNP levels at 12 months from baseline in both Treatment and Control groups during the overall follow-up period were analyzed using a mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 235 | 221
pg/mL | -80.61 (53.17) | -20.82 (55.51)
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group vs Randomized Arm - Control Group; Comparisons of change from baseline in BNP levels at 12 months between Treatment vs Control group; Test type: Superiority; p = 0.4373, Mixed Models Analysis; Least Square Means Difference (T vs C) = 59.78, 95% CI 2-sided [-91.44 to 211.01], Standard Error of Mean 76.87

60. Other Pre Specified Outcome: (Randomized Arm) NT-proBNP
Description: Change in NT-proBNP measurements from baseline
Time Frame: 6 months post-implantation
Population: Subjects that have a baseline value and at least one value at 6-month visit were analyzed. The Least Square Means (LSM) difference in NT-proBNP levels at 6 months from baseline in both Treatment and Control groups during the overall follow-up period were analyzed using a mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group
Number analyzed (Participants) | 184 | 193
pg/mL | -169.94 (183.37) | 298.16 (179.58)
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group vs Randomized Arm - Control Group; Comparisons of change from baseline in NT-proBNP levels at 6months between Treatment vs Control group; Test type: Superiority; p = 0.0692, Mixed Models Analysis; Least Square Means Difference (T vs C) = 468.10, 95% CI 2-sided [-37.09 to 973.30], Standard Error of Mean 256.65

61. Other Pre Specified Outcome: (Randomized Arm) NT-proBNP
Description: Change in NT-proBNP measurements from baseline
Time Frame: 12 months post-implantation
Population: Subjects that have a baseline value and at least one value at 12-month visit were analyzed. The Least Square Means (LSM) difference in NT-proBNP levels at 12 months from baseline in both Treatment and Control groups during the overall follow-up period were analyzed using a mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Randomized Arm - Treatment Group (12 Month) | Randomized Arm - Control Group (12 Month)
Number analyzed (Participants) | 184 | 193
pg/mL | 217.23 (190.28) | 501.90 (189.74)
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group (12 Month) vs Randomized Arm - Control Group (12 Month); Comparisons of change from baseline in NT-proBNP levels at 12 months between Treatment vs Control group; Test type: Superiority; p = 0.2903, Mixed Models Analysis; Least Square Means Difference (T vs C) = 284.67, 95% CI 2-sided [-244.27 to 813.60], Standard Error of Mean 268.72

62. Other Pre Specified Outcome: (Randomized Arm) HFHs Post- vs. Pre-implantation [Treatment Group]
Description: The number of HFHs at 12 months post-implantation compared to the number of HFHs in the 12 months prior to implantation in the Treatment group
Time Frame: 12 months post-implantation vs 12 months pre-implantation
Population: A comparison of HF hospitalizations in the 12 months prior to implantation compared to 12 months post implantation for the endpoint contributing population, which includes subjects of NYHA class II/III/IV with successful implantation and randomized into the Treatment group were analyzed.
Measure: Number; unit: events per patient-year
Groups:
- Randomized Arm - Treatment Group (One Year Prior to Implant); Randomized Arm - Treatment Group (One Year After Implant): Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Randomized Arm - Treatment Group (One Year Prior to Implant) | Randomized Arm - Treatment Group (One Year After Implant)
Number analyzed (Participants) | 497 | 497
events per patient-year | 0.643 | 0.415
Statistical Analysis 1: Comparison: Randomized Arm - Treatment Group (One Year Prior to Implant) vs Randomized Arm - Treatment Group (One Year After Implant); Test type: Superiority; p < 0.0001, Anderson-Gill model (robust sandwich); Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.53 to 0.78]

63. Other Pre Specified Outcome: (Randomized Arm) HFHs Post- vs. Pre-implantation [Control Group]
Description: The number of HFHs at 12 months post-implantation compared to the number of HFHs in the 12 months prior to implantation
Time Frame: 12 months post-implantation vs 12 months pre-implantation
Population: A comparison of HF hospitalizations in the 12 months prior to implantation compared to 12 months post implantation for the endpoint contributing population, which includes subjects of NYHA class II/III/IV with successful implantation and randomized into the Control group were analyzed.
Measure: Number; unit: events per patient-year
Groups:
- Randomized Arm - Control Group (One Year Prior to Implant); Randomized Arm - Control Group (One Year After Implant): Management of subjects per standard of care (signs, symptoms, weight etc.) without knowledge of PA pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Randomized Arm - Control Group (One Year Prior to Implant) | Randomized Arm - Control Group (One Year After Implant)
Number analyzed (Participants) | 503 | 503
events per patient-year | 0.710 | 0.483
Statistical Analysis 1: Comparison: Randomized Arm - Control Group (One Year Prior to Implant) vs Randomized Arm - Control Group (One Year After Implant); Test type: Superiority; p < 0.0001, Anderson-Gill model (robust sandwich); Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.57 to 0.81]

64. Other Pre Specified Outcome: (Single Arm) KCCQ-12 [Mixed Model Analysis]
Description: Health status as assessed by the KCCQ-12 The Kansas City Cardiomyopathy Questionnaire (KCCQ-12) is a validated health-related quality of life measure for heart failure and was qualified by the FDA as a medical device development tool in 2017. The KCCQ-12 quantifies physical function, symptoms (frequency, severity, and recent change), social function, self-efficacy and knowledge, and quality of life on a scale from 0 to 100. An overall summary score (OSS) is derived by averaging scores from each domain, with a higher score reflecting a better health status.
Time Frame: 6 months post-implantation
Population: The change in KCCQ-12 scores at 6 months visit from baseline in each qualification criteria group were analyzed using mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 423 | 506 | 290
scores on a scale | 6.19 (0.98) | 5.47 (0.90) | 10.70 (1.18)

65. Other Pre Specified Outcome: (Single Arm) KCCQ-12 [Mixed Model Analysis]
Description: as for outcome 64
Time Frame: 12 months post-implantation
Population: The change in KCCQ-12 scores at 12 months visit from baseline in each qualification criteria group were analyzed using mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 379 | 437 | 245
scores on a scale | 6.53 (1.07) | 5.00 (0.99) | 11.85 (1.32)

66. Other Pre Specified Outcome: (Single Arm) EQ-5D-5L [Mixed Model Analysis]
Description: Health status as assessed by the EQ-5D-5L Questionnaire. The data represents the EQ Visual Analogue Scale (VAS) subscale. The VAS records the subject's self-rated health status which ranges from a score of 0 (worst health you can imagine) to 100 (best health you can imagine). A higher VAS score for represents a better quality of life.
Time Frame: 6 months post-implantation
Population: The EQ-5D-5L scores at 6-month visit from baseline for each qualification criteria group were compared using Mixed Model Analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 423 | 506 | 292
scores on a scale | 3.86 (0.91) | 3.05 (0.83) | 2.41 (1.09)

67. Other Pre Specified Outcome: (Single Arm) EQ-5D-5L [Mixed Model Analysis]
Description: as for outcome 66
Time Frame: 12 months post-implantation
Population: The EQ-5D-5L scores at 12-month visit from baseline for each qualification criteria group were compared using Mixed Model Analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 379 | 437 | 246
scores on a scale | 3.42 (0.94) | 0.83 (0.88) | 4.93 (1.16)

68. Other Pre Specified Outcome: (Single Arm) 6MHW Test [Mixed Model Analysis]
Description: 6MHW Test Distance
Time Frame: 6 months post-implantation
Population: The 6MHW distance at 6 months from baseline in each qualification criteria group were compared using mixed model analysis. Subjects who were unable to walk due to heart failure symptoms were assigned zero meters.
Measure: Least Squares Mean (Standard Error); unit: meters, m
Groups:
- Single Arm - Elevated NT-proBNP/BNP Only [6 Month]: All subjects had prior elevated NT-proBNP/BNP only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm - Previous HF Hospitalization Only [6 Month]: All subjects had prior HF hospitalization only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [6 Month]: All subjects had prior elevated NT-proBNP/BNP and HF hospitalization with successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [6 Month] | Single Arm - Previous HF Hospitalization Only [6 Month] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [6 Month]
Number analyzed (Participants) | 429 | 503 | 314
meters, m | 5.25 (5.40) | 0.67 (5.13) | 20.11 (6.62)

69. Other Pre Specified Outcome: (Single Arm) 6MHW Test [Mixed Model Analysis]
Description: 6MHW Test Distance
Time Frame: 12 months post-implantation
Population: The 6MHW distance at 12 months from baseline in each qualification criteria group were compared using mixed model analysis. Subjects who were unable to walk due to heart failure symptoms were assigned zero meters.
Measure: Least Squares Mean (Standard Error); unit: meters, m
Groups:
- Single Arm - Elevated NT-proBNP/BNP Only [12 Month]: All subjects had prior elevated NT-proBNP/BNP only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm - Previous HF Hospitalization Only [12 Month]: All subjects had prior HF hospitalization only and successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
- Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [12 Month]: All subjects had prior elevated NT-proBNP/BNP and HF hospitalization with successful implant of CardioMEMS™ HF System.
  Management of subjects based on PA pressure information derived from the CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [12 Month] | Single Arm - Previous HF Hospitalization Only [12 Month] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [12 Month]
Number analyzed (Participants) | 429 | 503 | 314
meters, m | -3.80 (5.90) | -5.56 (5.99) | 20.18 (7.67)

70. Other Pre Specified Outcome: (Single Arm) Cardiovascular Mortality
Description: The number of deaths of cardiovascular cause
Time Frame: 12 months post-implantation
Population: The number of deaths that were cardiovascular in nature were analyzed in all three qualification criteria groups.
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 549 | 343
events per patient-year | 0.073 | 0.090 | 0.163

71. Other Pre Specified Outcome: (Single Arm) All-cause Hospitalizations
Description: The number of hospitalizations of any cause
Time Frame: 12 months post-implantation
Population: All-cause hospitalizations (overnight hospitalizations for any reason, including HF) were analyzed in all three qualification criteria groups.
Measure: Number; unit: events per patient-year
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 549 | 343
events per patient-year | 0.80 | 1.216 | 1.503

72. Other Pre Specified Outcome: (Single Arm) Frequency of Subject PA Pressure Uploads - Daily Compliance
Description: The frequency of subject uploads of PA pressure
Time Frame: 12 months post-implantation
Population: Subjects with at least one eligible day during the analysis period are included in the analysis. The daily compliance (percentage of eligible days in which a subject had a reading) per subject were analyzed in the endpoint contributing population that had at least one reading post-discharge from the implantation. Days when subjects did not have any reading taken during the eligible days are counted as zeroes.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 548 | 342
Percentage | 79 (22) | 72 (27) | 74 (25)

73. Other Pre Specified Outcome: (Single Arm) Frequency of Subject PA Pressure Uploads - Weekly Compliance
Description: The frequency of subject uploads of PA pressure
Time Frame: 12 months post-implantation
Population: Subjects with at least one eligible day during the analysis period are included in the analysis. The weekly compliance (percentage of weeks in which a subject had at least one reading) per subject were analyzed in the endpoint contributing population that had at least one reading post-discharge from the implantation. A week is considered eligible if the subject was eligible for readings three or more days during that week.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 546 | 342
Percentage | 0.94 (0.14) | 0.90 (0.20) | 0.91 (0.17)

74. Other Pre Specified Outcome: (Single Arm) HF Medication Changes
Description: The number of changes in HF medications
Time Frame: 12 months post-implantation
Population: The number of subjects with medication changes and the total number of medications changes are provided below for different classes of HF medications for each qualification criteria group.
Measure: Number; unit: Number of events
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 549 | 343
Number of events
  Diuretics: number analyzed (Participants) | 321 | 392 | 266
  Diuretics | 3026 | 4573 | 2630
  Angiotensin-Converting Enzyme (ACE) Inhibitors: number analyzed (Participants) | 30 | 35 | 20
  Angiotensin-Converting Enzyme (ACE) Inhibitors | 50 | 69 | 42
  Angiotensin Receptor Blocker (ARB): number analyzed (Participants) | 37 | 56 | 29
  Angiotensin Receptor Blocker (ARB) | 61 | 127 | 57
  Angiotensin Receptor-Neprilysin Inhibitor (ARNi): number analyzed (Participants) | 71 | 52 | 47
  Angiotensin Receptor-Neprilysin Inhibitor (ARNi) | 122 | 135 | 98
  Beta Blockers: number analyzed (Participants) | 132 | 161 | 113
  Beta Blockers | 285 | 358 | 239
  Mineralocorticoid Receptor Antagonist: number analyzed (Participants) | 99 | 159 | 95
  Mineralocorticoid Receptor Antagonist | 238 | 409 | 216
  SGLT2 Inhibitor: number analyzed (Participants) | 46 | 45 | 29
  SGLT2 Inhibitor | 73 | 66 | 46
  Nitrates: number analyzed (Participants) | 35 | 51 | 38
  Nitrates | 68 | 88 | 68
  Hydralazine/Other Vasodilators: number analyzed (Participants) | 37 | 57 | 43
  Hydralazine/Other Vasodilators | 93 | 121 | 102
  Calcium Channel Blockers: number analyzed (Participants) | 31 | 52 | 29
  Calcium Channel Blockers | 48 | 82 | 48
  Digoxin: number analyzed (Participants) | 21 | 16 | 9
  Digoxin | 37 | 23 | 18
  Sinus Node If Channel Inhibitors: number analyzed (Participants) | 2 | 2 | 1
  Sinus Node If Channel Inhibitors | 2 | 3 | 1

75. Other Pre Specified Outcome: (Single Arm) PA Pressure Measurements [Mixed Model Analysis]
Description: as for outcome 56
Time Frame: Baseline through 12 months post-implantation
Population: Change in PA pressure at 6 and 12 month visits from baseline was analyzed in each qualification group using a mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only [6 Month] | Single Arm - Previous HF Hospitalization Only [6 Month] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [6 Month] | Single Arm - Elevated NT-proBNP/BNP Only [12 Month] | Single Arm - Previous HF Hospitalization Only [12 Month] | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization [12 Month]
Number analyzed (Participants) | 416 | 496 | 286 | 357 | 399 | 233
mmHg
  Change in PA Systolic Pressure | -3.79 (0.43) | -3.32 (0.39) | -3.86 (0.52) | -3.49 (0.49) | -3.34 (0.46) | -4.32 (0.60)
  Change in PA Diastolic Pressure | -2.93 (0.26) | -2.34 (0.24) | -2.66 (0.31) | -2.71 (0.29) | -2.57 (0.27) | -3.17 (0.36)
  Change in PA Mean Pressure | -3.22 (0.32) | -2.73 (0.29) | -3.07 (0.39) | -2.92 (0.36) | -2.84 (0.34) | -3.60 (0.44)

76. Other Pre Specified Outcome: (Single Arm) PA Pressure Measurements [AUC Analysis]
Description: Changes in PA pressure relative to baseline for systolic, diastolic, and mean PA pressures analyzed using area under the curve (AUC) analysis of PA pressure across the full follow-up period
Time Frame: Baseline through 12 months post-implantation
Population: Change in PA pressure at 6 and 12 month visits from baseline were analyzed in each qualification group using AUC analysis.
Measure: Mean (Standard Deviation); unit: mmHg*Days
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 549 | 343
mmHg*Days
  PA Systolic Pressure: number analyzed (Participants) | 321 | 360 | 194
  PA Systolic Pressure | -1033.79 (2457.95) | -1021.13 (2374.17) | -1179.42 (2588.90)
  PA Diastolic Pressure: number analyzed (Participants) | 321 | 360 | 194
  PA Diastolic Pressure | -868.16 (1410.07) | -723.29 (1529.73) | -847.94 (1489.96)
  PA Mean Pressure: number analyzed (Participants) | 321 | 360 | 194
  PA Mean Pressure | -929.39 (1794.20) | -832.21 (1832.20) | -973.97 (1904.05)

77. Other Pre Specified Outcome: (Single Arm) NT-proBNP (or BNP) [Mixed Model Analysis]
Description: Either change in N-terminal pro-brain natriuretic peptide (NT-proBNP) or Brain natriuretic peptide (BNP) measurements at 6 months visits from baseline.
Time Frame: 6 months post-implantation
Population: Either BNP or NT-proBNP levels were measured at baseline, 6 months and 12 months in each qualification criteria group. Change from baseline at 6 months were analyzed using mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 549 | 343
pg/mL
  BNP: number analyzed (Participants) | 177 | 246 | 143
  BNP | 40.81 (38.50) | -103.33 (32.91) | -6.45 (41.50)
  NT-proBNP: number analyzed (Participants) | 214 | 224 | 125
  NT-proBNP | -55.40 (153.36) | -174.83 (151.97) | -102.91 (194.87)

78. Other Pre Specified Outcome: (Single Arm) NT-proBNP (or BNP) [Mixed Model Analysis]
Description: Either change in N-terminal pro-brain natriuretic peptide (NT-proBNP) or Brain natriuretic peptide (BNP) measurements at 6 months and 12 months visits from baseline.
Time Frame: 12 months post-implantation
Population: Either BNP or NT-proBNP levels were measured at baseline, 6 months and 12 months in each qualification criteria group. Change from baseline at 12 months were analyzed using mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Single Arm - Elevated NT-proBNP/BNP Only | Single Arm - Previous HF Hospitalization Only | Single Arm - Elevated NT-proBNP/BNP and Previous HF Hospitalization
Number analyzed (Participants) | 452 | 549 | 343
pg/mL
  BNP: number analyzed (Participants) | 161 | 221 | 129
  BNP | -11.23 (37.73) | -79.01 (32.23) | -17.71 (41.92)
  NT-proBNP: number analyzed (Participants) | 195 | 200 | 106
  NT-proBNP | -15.17 (206.01) | 348.49 (214.19) | 259.33 (279.57)

ADVERSE EVENTS:
Time Frame: Adverse device effects (ADEs), serious adverse device effects (SADEs), serious adverse events (SAEs), and unanticipated adverse device effects (UADEs) were summarized for subjects enrolled in this trial as number of events, the number and percentage of subjects with events and event rate as number of events/subject-month. Adverse event data were collected during the 1-year follow-up period.
Description: Serious Adverse Events listed below are either device-related (SADEs) or non-device related (SAEs), as denoted by the numbered subscripts. No UADEs were reported in the Randomized Arm and Single Arm adjudicated as such by the Clinical Events Committee (CEC).
Groups:
- Single Arm: Management of subjects based on pulmonary artery (PA) pressure information derived from the CardioMEMS™ HF System.
  All subjects will receive a CardioMEMS™ HF System.
  CardioMEMS™ HF System: The CardioMEMS™ HF System is comprised of a lead-less, battery-less pressure sensor permanently implanted in the PA, which remotely transmits PA pressure measurements from the patient's home to a secure website. Healthcare professionals are able to access these measurements and associated waveforms to remotely guide individualization of medical management for their patients with chronic HF.
  Total efficacy population includes implanted subjects not belonging to a qualifying group.
Arm/Group | Randomized Arm - Treatment Group | Randomized Arm - Control Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 40/497 | 37/503 | 190/1358
Serious Adverse Events (participants affected / at risk) | 283/497 | 272/503 | 820/1358
Other Adverse Events (participants affected / at risk) | 15/497 | 20/503 | 33/1358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Arm - Treatment Group (N=497) | Randomized Arm - Control Group (N=503) | Single Arm (N=1358)
Anemia (Blood and lymphatic system disorders) | 6 (9) | 7 (8) | 33 (41) — Non-device-related serious adverse events (SAEs)
Hemorrhagic Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Splenic Infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Angina Pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 3 (4) — Non-device-related serious adverse events (SAEs)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1) | 4 (5) — Non-device-related serious adverse events (SAEs)
Aortic Valve Disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Arrhythmia (Cardiac disorders) | 47 (53) | 46 (54) | 138 (158) — Non-device-related serious adverse events (SAEs)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) — Serious Adverse Device Affects (SADEs)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Cardiac Aneurysm (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Cardiac Arrest (Cardiac disorders) | 3 (3) | 4 (4) | 11 (11) — Non-device-related serious adverse events (SAEs)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Cardiac Failure Chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Cardiac Failure Congestive (Cardiac disorders) | 130 (216) | 155 (276) | 454 (776) — Non-device-related serious adverse events (SAEs)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) — Serious Adverse Device Affects (SADEs)
Cardiac Perforation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Cardiac Pseudoaneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Cardiac Tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Cardiac Valve Disease (Cardiac disorders) | 1 (1) | 3 (4) | 0 (0) — Non-device-related serious adverse events (SAEs)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Cardiogenic Shock (Cardiac disorders) | 8 (8) | 5 (6) | 10 (10) — Non-device-related serious adverse events (SAEs)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Cardiorenal Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 8 (9) | 9 (9) — Non-device-related serious adverse events (SAEs)
Hypertensive Heart Disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Intracardiac Thrombus (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Ischemic Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Mitral Valve Disease (Cardiac disorders) | 1 (1) | 2 (3) | 2 (2) — Non-device-related serious adverse events (SAEs)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Myocardial Infarction (Cardiac disorders) | 10 (11) | 16 (16) | 30 (32) — Non-device-related serious adverse events (SAEs)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Serious Adverse Device Affects (SADEs)
Myocardial Ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) — Non-device-related serious adverse events (SAEs)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Prinzmetal Angina (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) — Non-device-related serious adverse events (SAEs)
Restrictive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Right Ventricular Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 3 (3) — Non-device-related serious adverse events (SAEs)
Shone Complex (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) — Non-device-related serious adverse events (SAEs)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Colitis Ischemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Colonic Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (5) — Non-device-related serious adverse events (SAEs)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6) — Non-device-related serious adverse events (SAEs)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Enterocutaneous Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Esophageal Achalasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Esophageal Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) — Non-device-related serious adverse events (SAEs)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Gastritis Hemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 9 (10) | 16 (20) | 52 (64) — Non-device-related serious adverse events (SAEs)
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Intestinal Ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Pancreatic Mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Pneumatosis Intestinalis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Retroperitoneal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 9 (12) — Non-device-related serious adverse events (SAEs)
Spigelian Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) — Non-device-related serious adverse events (SAEs)
Accidental Death (General disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Adverse Drug Reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Asthenia (General disorders) | 4 (4) | 3 (3) | 11 (11) — Non-device-related serious adverse events (SAEs)
Catheter Site Hematoma (General disorders) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Catheter Site Hematoma (General disorders) | 0 (0) | 1 (1) | 2 (2) — Serious Adverse Device Affects (SADEs)
Catheter Site Hemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Catheter Site Hemorrhage (General disorders) | 4 (4) | 1 (1) | 2 (2) — Serious Adverse Device Affects (SADEs)
Chest Pain (General disorders) | 27 (32) | 23 (25) | 32 (36) — Non-device-related serious adverse events (SAEs)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) — Serious Adverse Device Affects (SADEs)
Device Deployment Issue (General disorders) | 0 (0) | 1 (1) | 0 (0) — Serious Adverse Device Affects (SADEs)
Device Dislocation (General disorders) | 2 (2) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Device Dislocation (General disorders) | 0 (0) | 1 (1) | 1 (1) — Serious Adverse Device Affects (SADEs)
Device Electrical Impedance Issue (General disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Device Information Output Issue (General disorders) | 0 (0) | 0 (0) | 1 (1) — Serious Adverse Device Affects (SADEs)
Device malfunction (General disorders) | 0 (0) | 3 (3) | 3 (3) — Non-device-related serious adverse events (SAEs)
Edema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Generalized Edema (General disorders) | 1 (2) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Impaired Healing (General disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Implant Site Hemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Multi-Organ Failure (General disorders) | 1 (1) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 25 (26) — Non-device-related serious adverse events (SAEs)
Polyp (General disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Sudden Cardiac Death (General disorders) | 1 (1) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Systemic Inflammatory Response Syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Thrombosis In Device (General disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Ulcer (General disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Unintentional Medical Device Removal By Patient (General disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Unknown Event Leading to Death (General disorders) | 3 (3) | 0 (0) | 11 (11) — Non-device-related serious adverse events (SAEs)
Unknown Event Leading to Death (General disorders) | 0 (0) | 0 (0) | 3 (3) — Serious Adverse Device Affects (SADEs)
Acute Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Bile Duct Stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Cardiac Cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2) — Non-device-related serious adverse events (SAEs)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Hepatic Cirrhosis (Hepatobiliary disorders) | 2 (2) | 2 (2) | 3 (3) — Non-device-related serious adverse events (SAEs)
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Hepatitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Ischemic Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Heart Transplant Rejection (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Abdominal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Anal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Bronchitis (Infections and infestations) | 2 (2) | 7 (7) | 5 (5) — Non-device-related serious adverse events (SAEs)
Cellulitis (Infections and infestations) | 5 (6) | 7 (8) | 8 (8) — Non-device-related serious adverse events (SAEs)
Central Nervous System Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Chest Wall Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Clostridial Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Corona Virus Infection (Infections and infestations) | 1 (1) | 2 (2) | 27 (31) — Non-device-related serious adverse events (SAEs)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) — Non-device-related serious adverse events (SAEs)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Gastrointestinal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Implant Site Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Infection (Infections and infestations) | 27 (29) | 34 (39) | 103 (119) — Non-device-related serious adverse events (SAEs)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Intervertebral Discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Mycotic Aneurysm (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Perineal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Pneumonia (Infections and infestations) | 24 (27) | 29 (32) | 71 (78) — Non-device-related serious adverse events (SAEs)
Pneumonia Parainfluenza Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Pneumonia Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Rocky Mountain Spotted Fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Sepsis (Infections and infestations) | 17 (18) | 10 (10) | 48 (57) — Non-device-related serious adverse events (SAEs)
Septic Shock (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) — Non-device-related serious adverse events (SAEs)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) — Non-device-related serious adverse events (SAEs)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 4 (4) | 9 (10) — Non-device-related serious adverse events (SAEs)
Vestibular Neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Arterial Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) — Serious Adverse Device Affects (SADEs)
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 17 (18) | 13 (17) | 43 (51) — Non-device-related serious adverse events (SAEs)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 5 (6) | 17 (17) — Non-device-related serious adverse events (SAEs)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 5 (5) — Non-device-related serious adverse events (SAEs)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Gastrointestinal Disorder Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Hip Fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 6 (6) — Non-device-related serious adverse events (SAEs)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Iliotibial Band Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Open Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) — Non-device-related serious adverse events (SAEs)
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Post Procedural Hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Post Procedural Oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Snake Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (3) — Non-device-related serious adverse events (SAEs)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) — Non-device-related serious adverse events (SAEs)
Sternal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Subdural Hematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 6 (6) — Non-device-related serious adverse events (SAEs)
Tendon Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Traumatic Arthropathy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Traumatic Intracranial Hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Vaccination Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) — Serious Adverse Device Affects (SADEs)
Anticoagulation Drug Level Below Therapeutic (Investigations) | 1 (1) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Blood Magnesium Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Device Function Test (Investigations) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
International Normalized Ratio Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
International Normalized Ratio Increased (Investigations) | 0 (0) | 1 (1) | 4 (4) — Non-device-related serious adverse events (SAEs)
Left Ventricular End-Diastolic Pressure Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Transaminases Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Troponin Increased (Investigations) | 1 (1) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 2 (2) | 12 (13) — Non-device-related serious adverse events (SAEs)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 7 (7) — Non-device-related serious adverse events (SAEs)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Fluid Overload (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 2 (3) — Non-device-related serious adverse events (SAEs)
Gout (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 7 (9) — Non-device-related serious adverse events (SAEs)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5) | 4 (5) | 14 (15) — Non-device-related serious adverse events (SAEs)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Serious Adverse Device Affects (SADEs)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 15 (17) — Non-device-related serious adverse events (SAEs)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 6 (6) — Non-device-related serious adverse events (SAEs)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 9 (12) — Non-device-related serious adverse events (SAEs)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (8) — Non-device-related serious adverse events (SAEs)
Hypovolemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (2) — Non-device-related serious adverse events (SAEs)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Lactic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 6 (6) — Non-device-related serious adverse events (SAEs)
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Serious Adverse Device Affects (SADEs)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) — Non-device-related serious adverse events (SAEs)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Biliary Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Esophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3) — Non-device-related serious adverse events (SAEs)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Mantle Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 4 (5) — Non-device-related serious adverse events (SAEs)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Small Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
CNS Ventriculitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) — Non-device-related serious adverse events (SAEs)
Cerebral Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Cerebrovascular Accident (Nervous system disorders) | 11 (12) | 6 (6) | 15 (16) — Non-device-related serious adverse events (SAEs)
Cerebrovascular Disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Cervical Cord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Cervicogenic Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Complicated Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) — Non-device-related serious adverse events (SAEs)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Dementia with Lewy Bodies (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Diabetic Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4) | 6 (6) — Non-device-related serious adverse events (SAEs)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 6 (7) — Non-device-related serious adverse events (SAEs)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Hemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Hepatic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) — Non-device-related serious adverse events (SAEs)
Hypoesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
IIIrd (Third) Nerve Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Metabolic Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) — Non-device-related serious adverse events (SAEs)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Orthostatic Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Partial Seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Presyncope (Nervous system disorders) | 3 (3) | 0 (0) | 3 (4) — Non-device-related serious adverse events (SAEs)
Renal Failure (Nervous system disorders) | 3 (3) | 1 (1) | 8 (8) — Non-device-related serious adverse events (SAEs)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Subarachnoid Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Syncope (Nervous system disorders) | 12 (12) | 8 (8) | 24 (24) — Non-device-related serious adverse events (SAEs)
Transient Ischemic Attack (Nervous system disorders) | 2 (2) | 0 (0) | 8 (9) — Non-device-related serious adverse events (SAEs)
Vascular Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Vertebral Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Serious Adverse Device Affects (SADEs)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (4) — Non-device-related serious adverse events (SAEs)
Depression (Psychiatric disorders) | 0 (0) | 2 (3) | 1 (1) — Non-device-related serious adverse events (SAEs)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Mental Status Changes (Psychiatric disorders) | 2 (2) | 3 (3) | 8 (8) — Non-device-related serious adverse events (SAEs)
Azotemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Calculus Ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 4 (4) — Non-device-related serious adverse events (SAEs)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) — Non-device-related serious adverse events (SAEs)
Obstructive Uropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Renal Failure Acute (Renal and urinary disorders) | 18 (21) | 28 (29) | 81 (95) — Non-device-related serious adverse events (SAEs)
Renal Failure Chronic (Renal and urinary disorders) | 2 (2) | 5 (6) | 3 (3) — Non-device-related serious adverse events (SAEs)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Renal Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Urinary Retention (Renal and urinary disorders) | 3 (3) | 2 (2) | 1 (1) — Non-device-related serious adverse events (SAEs)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Uterovaginal Prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8) | 26 (28) — Non-device-related serious adverse events (SAEs)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 14 (24) | 37 (48) — Non-device-related serious adverse events (SAEs)
Chronic Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Non-device-related serious adverse events (SAEs)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (8) | 7 (8) — Non-device-related serious adverse events (SAEs)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 5 (6) — Non-device-related serious adverse events (SAEs)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4) — Non-device-related serious adverse events (SAEs)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2) — Serious Adverse Device Affects (SADEs)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Laryngeal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4) | 5 (5) — Non-device-related serious adverse events (SAEs)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) — Non-device-related serious adverse events (SAEs)
Pulmonary Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) — Serious Adverse Device Affects (SADEs)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (3) — Non-device-related serious adverse events (SAEs)
Pulmonary Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 6 (7) — Non-device-related serious adverse events (SAEs)
Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) — Non-device-related serious adverse events (SAEs)
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) — Non-device-related serious adverse events (SAEs)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Substance Use (Social circumstances) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Aneurysm (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Aortic Valve Replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Cardiac Pacemaker Battery Replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Cardiac Pacemaker Replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) — Non-device-related serious adverse events (SAEs)
Implantable Defibrillator Insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Aortic Aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Aortic Stenosis (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) — Non-device-related serious adverse events (SAEs)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Bleeding Varicose Vein (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Blood Pressure Fluctuation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Embolism (Vascular disorders) | 2 (2) | 0 (0) | 5 (5) — Non-device-related serious adverse events (SAEs)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — Serious Adverse Device Affects (SADEs)
Extremity Necrosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Hematoma (Vascular disorders) | 2 (2) | 0 (0) | 9 (10) — Non-device-related serious adverse events (SAEs)
Hematoma (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) — Serious Adverse Device Affects (SADEs)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) — Non-device-related serious adverse events (SAEs)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 2 (2) | 2 (2) — Non-device-related serious adverse events (SAEs)
Hypertensive Emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Hypotension (Vascular disorders) | 13 (14) | 11 (11) | 34 (34) — Non-device-related serious adverse events (SAEs)
Hypovolemic Shock (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) — Non-device-related serious adverse events (SAEs)
Lymphoedema (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) — Non-device-related serious adverse events (SAEs)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 6 (7) — Non-device-related serious adverse events (SAEs)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1) | 2 (2) | 7 (7) — Non-device-related serious adverse events (SAEs)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Shock Hemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) — Non-device-related serious adverse events (SAEs)
Subclavian Artery Stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Thrombosis (Vascular disorders) | 4 (5) | 2 (3) | 6 (6) — Non-device-related serious adverse events (SAEs)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) — Serious Adverse Device Affects (SADEs)
Varicose Ulceration (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Venous Insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Non-device-related serious adverse events (SAEs)
Vessel Perforation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Serious Adverse Device Affects (SADEs)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Arm - Treatment Group (N=497) | Randomized Arm - Control Group (N=503) | Single Arm (N=1358)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2) | 3 (3) — Non-serious Adverse Device Effects (ADEs)
Catheter Site Hematoma (General disorders) | 2 (2) | 3 (3) | 2 (2) — Non-serious Adverse Device Effects (ADEs)
Catheter Site Hemorrhage (General disorders) | 4 (4) | 6 (6) | 10 (10) — Non-serious Adverse Device Effects (ADEs)
Device Deployment Issue (General disorders) | 0 (0) | 1 (1) | 1 (1) — Non-serious Adverse Device Effects (ADEs)
Device Dislocation (General disorders) | 0 (0) | 3 (3) | 7 (7) — Non-serious Adverse Device Effects (ADEs)
Device Information Output Issue (General disorders) | 2 (2) | 2 (2) | 0 (0) — Non-serious Adverse Device Effects (ADEs)
Device Malfunction (General disorders) | 0 (0) | 1 (1) | 2 (2) — Non-serious Adverse Device Effects (ADEs)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) — Non-serious Adverse Device Effects (ADEs)
Vessel Puncture Site Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) — Non-serious Adverse Device Effects (ADEs)
Arterial Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Non-serious Adverse Device Effects (ADEs)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Non-serious Adverse Device Effects (ADEs)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) — Non-serious Adverse Device Effects (ADEs)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) — Non-serious Adverse Device Effects (ADEs)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) — Non-serious Adverse Device Effects (ADEs)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Non-serious Adverse Device Effects (ADEs)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Non-serious Adverse Device Effects (ADEs)
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-serious Adverse Device Effects (ADEs)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Non-serious Adverse Device Effects (ADEs)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Non-serious Adverse Device Effects (ADEs)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Non-serious Adverse Device Effects (ADEs)
Catheter Site Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) — Non-serious Adverse Device Effects (ADEs)

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic affected the GUIDE-HF Randomized Arm study. The impact of COVID-19 on the primary endpoint and components was addressed through sensitivity analyses.

Single Arm Total Efficacy Population includes implanted subjects not belonging to a qualifying criteria group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT03387813/Prot_002.pdf
  • Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT03387813/SAP_003.pdf